CLINICAL TRIAL: NCT02609828
Title: A PHASE 3 RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED, MULTICENTER STUDY OF THE ANALGESIC EFFICACY AND SAFETY OF THE SUBCUTANEOUS ADMINISTRATION OF TANEZUMAB (PF-04383119) IN SUBJECTS WITH CANCER PAIN PREDOMINANTLY DUE TO BONE METASTASIS RECEIVING BACKGROUND OPIOID THERAPY
Brief Title: Phase 3 Study on the Efficacy and Safety of Tanezumab in Patients With Cancer Pain Due to Bone Metastasis Who Are Taking Background Opioid Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A4091061; 2013-002223-42 (EudraCT Number); CANCER PAIN PH 3 SC STUDY (Other: Alias Study Number)
Record Dates: First submitted 2015-10-26; First posted 2015-11-20 (Estimated); Results first posted 2023-01-20 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-01

CONDITIONS: Bone Metastasis; Cancer Pain
Keywords: Metastatic cancer bone pain; Multiple myeloma
MeSH Terms: conditions — Cancer Pain; Multiple Myeloma | interventions — tanezumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Tanezumab 20 mg subcutaneously
  Interventions: Drug: Tanezumab
- Arm 2 (Placebo Comparator): Placebo matched to active treatment subcutaneously
  Interventions: Drug: Tanezumab

INTERVENTIONS:
Drug: Tanezumab — Subcutaneous study treatment (tanezumab 20 mg or matched placebo) dosed at 8 week intervals.
  Other Names: PF-04383119

SUMMARY:
The purpose of this study is to determine whether tanezumab is effective in the treatment of cancer pain due to bone metastasis in patients already taking background opioid therapy.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, multicenter, parallel-group Phase 3 study in cancer subjects requiring treatment with background opioids for pain due to bone metastasis.

Approximately 144 subjects will be randomized to one of 2 treatment groups in a 1:1 ratio (approximately 72 subjects per group). Subjects will receive a total of 3 subcutaneous injections, separated by 8 weeks in addition to background opioids administered throughout the study.

Treatment groups will include: 1. Placebo SC (matching tanezumab SC) in addition to background opioid therapy. 2. Tanezumab 20 mg SC in addition to background opioid therapy.

The study consists of three periods: Pre-Treatment (up to 37 days), Double-Blind Treatment (24 weeks) and Safety Follow-up (24 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Personally signed and dated informed consent document.
* Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
* Male or female, ≥18 years of age
* Weight ≥40 kg at Screening
* Cancer diagnosed as having metastasized to bone or multiple myeloma.
* Imaging confirmation of bone metastasis at Screening or within 120 days prior to the Screening visit.
* Expected to require daily opioid medication throughout the course of the study.
* Willing to not use prohibited medications (including NSAIDs) throughout the duration of the study.
* Average Pain Score ≥5 at Screening for the index bone metastasis cancer pain site.
* Patient's Global Assessment of Cancer Pain of "fair", "poor" or "very poor" at Screening.
* Eastern Cooperative Oncology Group (ECOG) Performance Status Score of 0, 1, or 2 at Screening.
* Adequate bone marrow, renal and liver function at Screening.
* International Normalized Ratio (INR) or prothrombin time (PT) <1.5 x ULN at Screening unless being treated with anticoagulant medication.
* Females must either be not of childbearing potential or, if of childbearing potential and at risk for pregnancy, must be willing to use at least one highly effective method of contraception throughout the study and for 112 days (16 weeks) after the last dose of assigned subcutaneous study medication.

Exclusion Criteria:

* Pain related to an oncologic emergency.
* Brain metastasis or leptomeningeal metastasis.
* Presence of hypercalcemia at Screening.
* Pain primarily classified as not predominantly related to a bone metastasis.
* Systemic treatment for the primary malignancy or bone metastasis started within 30 days of the Baseline Assessment Period.
* Chemotherapies associated with peripheral neuropathy (ie, paclitaxel, docetaxel, oxaliplatin, cisplatin, vincristine, thalidomide or bortezomib) are prohibited during the study from 30 days prior to the first day of the Baseline Assessment Period to Week 48.
* Receipt of radiopharmaceutical treatment or radiotherapy for treatment of bone metastasis within 30 days of the Baseline Assessment Period.
* Concurrent adjuvant analgesics unless started at least 30 days prior to the start of the Baseline Assessment Period and maintained at a stable dose.
* Diagnosis of osteoarthritis of the knee or hip or findings consistent with osteoarthritis in the shoulder.
* History of significant trauma or surgery to a major joint within one year prior to Screening.
* History of osteonecrosis or osteoporotic fracture.
* X-ray evidence at Screening of: 1) rapidly progressive osteoarthritis, 2) atrophic or hypotrophic osteoarthritis, 3) subchondral insufficiency fracture, 4) spontaneous osteonecrosis of the knee (SPONK), 5) osteonecrosis, or 6) pathologic fracture.
* Signs and symptoms of clinically significant cardiac disease.
* Evidence of orthostatic hypotension at Screening or at Baseline prior to randomization.
* Diagnosis of a transient ischemic attack in the 6 months prior to Screening or diagnosis of stroke with significant residual deficits.
* History, diagnosis, or signs and symptoms of clinically significant neurological disease.
* Total impact score of >7 on the Survey of Autonomic Symptoms (SAS) at Screening.
* Past history of carpal tunnel syndrome (CTS) with signs or symptoms of CTS in the one year prior to Screening.
* History of significant alcohol, analgesic, or narcotic substance abuse within the six months prior to Screening.
* Planned surgical procedure during the duration of the study.
* Considered unfit for surgery or not willing to undergo joint replacement surgery if required.
* Known hypersensitivity to opioids or an underlying medical condition contraindicating opioid use.
* History of allergic or anaphylactic reaction to a therapeutic or diagnostic monoclonal antibody or IgG-fusion protein.
* Previous exposure to exogenous nerve growth factor or to an anti-nerve growth factor antibody.
* Presence of drugs of abuse, prescription medications without a valid prescription or other illegal drugs at Screening.
* Positive Hepatitis B, Hepatitis C, or Human Immunodeficiency Virus (HIV) tests at Screening indicative of current infection.
* Investigational site staff members and their family members, or Pfizer employees directly involved in the conduct of the trial.
* Participation in other studies involving investigational drug(s) within 30 days (or 90 days for investigational biologics) before Baseline Assessment Period and/or during study participation.
* Pregnant female subjects; breastfeeding female subjects; female subjects of childbearing potential who are unwilling or unable to use one (1) highly effective method of contraception throughout the study and for 112 days after last dose of investigational product.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2015-10-28 (Actual); Primary Completion 2020-09-17 (Actual); Study Completion 2021-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (89):
- Instituto de Oncologia de Rosario, Rosario, Santa Fe Province, Argentina
- Australia (2):
  - Monash Medical Centre, Clayton, Victoria
  - Monash Medical Centre, East Bentleigh, Victoria
- Austria (2):
  - Landesklinikum Krems, Krems
  - Nuhr Medical Center, Senftenberg
- Brazil (10):
  - INCA - Instituto Nacional do Cancer / Hospital do Cancer HCIII, Rio de Janeiro, Rio de Janeiro
  - Associacao Hospital de Caridade de Ijui, Ijuí, Rio Grande do Sul
  - Centro de Novos Tratamentos Itajai - Clinica de Neoplasias Litoral, Itajaí, Santa Catarina
  - Fundação Pio XII-Hospital de Cancer de Barretos, Barretos, São Paulo
  - Centro de Ensino e Pesquisa da Fundacao Amaral Carvalho, Jaú, São Paulo
  - Fundacao do ABC - Faculdade de Medicina do ABC - CEPHO, Santo André, São Paulo
  - Fundacao do ABC-Faculdade de Medicina do ABC, Santo André, São Paulo
  - Hospital AC Camargo_Fundacao Antonio Prudente, São Paulo, São Paulo
  - Centro de Pesquisa Clinica do IBCC - Instituto Brasileiro de Controle do Cancer, São Paulo, São Paulo
  - Hospital AC Camargo_Fundacao Antonio Prudente, São Paulo
- James Lind Centro de lnvestigacion del Cancer, Araucania, Chile
- China (11):
  - The First Affiliated Hospital of Anhui Medical University, Department of Medical Oncology, Hefei, Anhui
  - The Fifth Medical Center of PLA General Hospital, Beijing, Beijing Municipality
  - Daping Hospital, Research Institute of Surgery Third Military Medical University, Chongqing, Chongqing Municipality
  - Harbin Medical University Cancer Hospital/Oncology Department, Harbin, Heilongjiang
  - Henan Cancer Hospital/Respiration internal medicine, Zhengzhou, Henan
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science & Technology/Cancer Center, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality
  - Oncology Department, West China Hospital of Sichuan University, Chengdu, Sichuan
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Tianjin Cancer Hospital, Tianjin
- Czechia (2):
  - Urocentrum Plzen Research Site s.r.o., Pilsen
  - Vseobecna fakultni nemocnice v Praze, Fakultni poliklinika, Centrum pro lecbu bolesti, Prague
- Hungary (6):
  - Veszprem Megyei Tudogyogyintezet Farkasgyepu, Farkasgyepű
  - CRU Hungary Ltd., MISEK Hematology Department-CRU Co., Miskolc
  - CRU Hungary Ltd., MISEK-CRU, Miskolc
  - Josa Andras Hospital, Clinical Research Department, Nyíregyháza
  - Szabolcs-Szatmar-Bereg Megyei Korhazak es Egyetemi Oktatokorhaz, Nyíregyháza
  - Help-MR Diagnosztika Kft., Székesfehérvár
- Israel (3):
  - HaEmek Medical Center, Afula
  - Rambam Health Care Campus, Haifa
  - Chaim Sheba Medical Center, Ramat Gan
- Japan (7):
  - National Hospital Organization Toyohashi Medical Center, Toyohashi, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Gunma Prefectural Cancer Center, Ōta, Gunma
  - Nishinomiya Municipal Central Hospital, Nishinomiya, Hyōgo
  - The Hospital of Hyogo College of Medicine, Nishinomiya, Hyōgo
  - Saga-Ken Medical Centre Koseikan, Saga
  - National Hospital Organization Tokyo Medical Center, Tokyo
- Poland (18):
  - Powiatowy Zespol Zakladow Opieki Zdrowotnej Oddzial Opieki Paliatywnej, Będzin
  - NZOZ Vitamed im. Edyty Jakubow, Bialystok
  - Poradnia Otropedyczno-Urazowa; Gabient RTG, Bialystok
  - Pracownia RTG Helimed, Czeladź
  - Niepubliczny Zaklad Opieki Zdrowotnej, Zespol Medyczno-Opiekunczy Alicja Kluczna, Dąbrowa Górnicza
  - Hospicjum im. Ks. Eugeniusza Dutkiewicza SAC w Gdansku, Gdansk
  - Stowarzyszenie Przyjaciol Chorych Hospicjum w Gliwicach NZOZ Hospicjum Milosierdzia Bozego, Gliwice
  - Stowarzyszenie Przyjaciol Chorych Hospicjum w Gliwicach, NZOZ Hospicjum Milosierdzia Bozego, Gliwice
  - Regionalny Szpital Specjalistyczny im. Dr. Wl.Bieganskiego, Oddzial Onkologii Klinicznej, Grudziądz
  - SCANiX Sp.z o.o, Katowice
  - NZOZ "Vegamed", Katowice
  - Helimed Diagnostic Imaging Sp. z o.o., Sp. komandytowa, Katowice
  - Helimed Diagnostic Imaging Sp. z.o.o., Sp. komandytowa, Katowice
  - Centrum Diagnostyki Obrazowej EPIONE, Katowice
  - NZOZ Neuromed M. i M. Nastaj Sp. P., Lublin
  - SK Przemienienia Panskiego UM im. Karola Marcinkowskiego w Poznaniu,, Poznan
  - Klinika Nowotworow Piersi i Chirurgii Rekonstrukcyjnej w Centrum Onkologii -Instytucie, Warsaw
  - Szpital LUX MED, Warsaw
- Romania (3):
  - SC Oncolab SRL, Craiova, Dolj
  - S.C. Oncocenter Oncologie Clinica S.R.L., Timișoara, Timiș County
  - Spitalul Clinic C.F. 2 Bucuresti. Departament Oncologie, Sectia Medicala 2, Bucharest
- Slovakia (4):
  - Narodny onkologicky ustav, Bratislava
  - DEMOMED s.r.o., Nové Zámky
  - MUDr. Viliam Cibik, PhD, s.r.o., Pruské
  - Fakultna Nemocnica S Poliklinikou Zilina, Žilina
- South Korea (8):
  - Clinical Trial Pharmacy, National Cancer Center, Goyang-si, Gyeonggi-do
  - Imaging Facilities, National Cancer Center, Goyang-si, Gyeonggi-do
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Keimyung University Dongsan Medical Center, Daegu
  - Clinical Trial Pharmacy, Severance Hospital, Seoul
  - Imaging Facilities, Severance Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
- Spain (7):
  - Hospital General Universitario de Elche Servicio de Farmacia, Elche, Alicante
  - Hospital General Universitario de Elche, Elche, Alicante
  - Hospital Can Misses, Ibiza Town, Balearic Islands
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitario de la Princesa, Madrid
  - Hospital La Moraleja, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
- United Kingdom (4):
  - St George's University Hospitals NHS Foundation Trust, Tooting, London
  - NHS Lothian, Royal Infirmary of Edinburgh, Edinburgh, Scotland
  - NHS Lothian, Western General Hospital, Edinburgh, Scotland
  - NHS Lothian, Edinburgh, Scotland

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Fallon M, Sopata M, Dragon E, Brown MT, Viktrup L, West CR, Bao W, Agyemang A. A Randomized Placebo-Controlled Trial of the Anti-Nerve Growth Factor Antibody Tanezumab in Subjects With Cancer Pain Due to Bone Metastasis. Oncologist. 2023 Dec 11;28(12):e1268-e1278. doi: 10.1093/oncolo/oyad188. PMID 37343145
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4091061&StudyName=A%20Phase%203%20Randomized%2C%20Double-blind%2C%20Placebo-controlled%2C%20Multicenter%20Study%20Of%20The%20Analgesic%20Efficacy%20And%20Safety%20Of%20The%20Subcutaneous%20Administration%20Of%20Tanezumab%20%28pf-04383119%29%20In%20Subjects%20With%20Cancer%20Pain%20Predominantly%20Due%20To%20Bone%20Metastasis%20Receiving%20Background%20Opioid%20Therapy

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with cancer pain predominantly due to bone metastasis and receiving background opioid therapy, were randomized into 3 treatment arms: tanezumab 20 milligrams (mg), tanezumab 10 mg and placebo. After study start, tanezumab 10 mg arm was discontinued in protocol amendment 3: no new participants were enrolled into the arm. Existing participants in the arm received tanezumab 20 mg for any remaining doses and were included in tanezumab 10/20 mg arm.
Pre-assignment Details: Total 325 participants signed the inform consent form (ICF). Out of which 158 participants were screen failures, and 11 participants were screened but not enrolled and randomized into the study. Total of 156 participants were enrolled and randomized into the study and assigned to study treatments.
Groups:
- Placebo: Participants received placebo matched to tanezumab subcutaneous (SC) once every 8 weeks for 24 weeks.
- Tanezumab 10 mg: Participants in this discontinued treatment arm, received tanezumab 10 mg SC once every 8 weeks before protocol amendment 3 and completed their treatment before the amendment.
- Tanezumab 10/20 mg: Participants in this treatment group had received tanezumab 10 mg SC once every 8 weeks before protocol amendment 3 and after the amendment they continued remaining treatment with tanezumab 20 mg SC once every 8 weeks.
- Tanezumab 20 mg: Participants received tanezumab 20 mg SC once every 8 weeks for 24 weeks.
Period: Overall Study
Arm/Group | Placebo | Tanezumab 10 mg | Tanezumab 10/20 mg | Tanezumab 20 mg
Started | 74 | 9 (A total of 10 participants were initially randomized to this arm. This arm was discontinued per protocol amendment 3. At time of amendment, out of 10 participants, 1 participant was still in treatment with tanezumab 10 mg. Post-amendment, this participant continued treatment with tanezumab 20 mg and was included in tanezumab 10/20 mg arm.) | 1 (The participant switched to this arm from tanezumab 10 mg post protocol amendment 3 implementation for remaining doses.) | 72
Treated | 73 | 9 | 1 | 72
Completed | 31 | 5 | 0 | 29
Not Completed | 43 | 4 | 1 | 43
Not completed — Adverse Event | 8 | 1 | 0 | 6
Not completed — Death | 15 | 1 | 1 | 19
Not completed — Insufficient clinical response | 2 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 2 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 12 | 1 | 0 | 10
Not completed — Other | 3 | 0 | 0 | 6
Not completed — Randomized but not treated | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants treated with tanezumab or placebo SC, including participants who received tanezumab 10 mg prior to protocol amendment 3.
Groups:
- Placebo: Participants received placebo matched to tanezumab SC once every 8 weeks for 24 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | Tanezumab 10 mg | Tanezumab 10/20 mg | Tanezumab 20 mg | Total
Number analyzed (Participants) | 73 | 9 | 1 | 72 | 155
Age, Customized [Count of Participants; unit: Participants]
  >=18 to <45 years | 10 | 1 | 0 | 3 | 14
  >=45 to <65 years | 44 | 4 | 1 | 33 | 82
  >=65 years | 19 | 4 | 0 | 36 | 59
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 4 | 0 | 26 | 69
  Male | 34 | 5 | 1 | 46 | 86
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 0 | 0 | 5 | 15
  Not Hispanic or Latino | 63 | 9 | 1 | 67 | 140
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 16 | 3 | 0 | 16 | 35
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1 | 2
  White | 56 | 6 | 1 | 55 | 118
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Daily Average Pain Intensity Numerical Rating Score (NRS) in the Index Bone Metastasis Cancer Pain Site at Week 8
Description: Daily average pain intensity in the index bone metastasis cancer pain site was assessed by participants on an 11 point pain intensity NRS ranging from 0 (no pain) to 10 (worst possible pain), where higher scores signified more severity of pain. The participants recorded their daily average pain at the painful site during the past 24 hours by choosing the appropriate number from 0 to 10 on interactive response technology (IRT) diaries. Baseline daily average pain intensity value was mean of the daily average pain intensity NRS scores during the baseline assessment period prior to randomization. Baseline assessment period was up to 5 days prior to dosing. The Week 8 daily average pain intensity value was the mean of the daily average pain intensity NRS scores recorded for each of the 7 days prior to the Week 8.
Time Frame: Baseline, Week 8
Population: The modified intent to treat (mITT) analysis set: participants randomized to tanezumab 20 mg or placebo SC, received at least 1dose of SC study medication. Multiple imputation method was applied. As planned summarized efficacy data for tanezumab 10 mg and 10/20 mg arms not reported; for these 2 arms individual values are reported. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Tanezumab 10 mg | Tanezumab 10/20 mg | Tanezumab 20 mg
Number analyzed (Participants) | 73 | 8 | 1 | 72
Units on a scale | -1.25 (0.35) | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual values were -3, -1.8, -0.6, -3.66, -2.4, -3, -1 and -2. | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual value was -0.48. | -2.03 (0.35)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 20 mg; Change at Week 8: Analysis of covariance (ANCOVA) model for imputed datasets included treatment, region, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness) as fixed effects, and baseline average pain intensity at the index bone metastasis cancer pain site and baseline opioid dose as covariates; Test type: Superiority; p = 0.0381, ANCOVA; Differences in least square (LS) mean = -0.78, 95% CI 2-sided [-1.52 to -0.04], Standard Error of Mean 0.37

2. Secondary Outcome: Change From Baseline in the Daily Average Pain Intensity NRS Score in the Index Bone Metastasis Cancer Pain Site at Weeks 1, 2, 4, 6, 12, 16 and 24
Description: Daily average pain intensity in the index bone metastasis cancer pain site was assessed by participants on an 11 point pain intensity NRS ranging from 0 (no pain) to 10 (worst possible pain) where higher scores signified more severity of pain. The participants recorded their daily average pain at the painful site during the past 24 hours by choosing the appropriate number from 0 to 10 on IRT diaries. Baseline daily average pain intensity value was mean of the daily average pain intensity NRS scores during the baseline assessment period prior to randomization. Baseline assessment period was up to 5 days prior to dosing. The Weeks 1, 2, 4, 6, 12, 16 and 24 daily average pain intensity value was the mean of the daily average pain intensity NRS scores recorded for each of the 7 days prior to the each specified week.
Time Frame: Baseline, Weeks 1, 2, 4, 6, 12, 16 and 24
Population: The mITT analysis set: participants randomized to tanezumab 20 mg or placebo SC, received at least 1dose of SC study medication. Multiple imputation method was applied. As planned summarized efficacy data for tanezumab 10 mg and 10/20 mg arms not reported; for these 2 arms individual values are reported. Here, ''number analyzed'' signifies participants evaluable at specified time points.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Tanezumab 10 mg | Tanezumab 10/20 mg | Tanezumab 20 mg
Number analyzed (Participants) | 73 | 9 | 1 | 72
Units on a scale
  Change at Week 1 | -0.40 (0.16) | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual values were 0, 0.2, -2.42, -0.45, -2.08, -0.4, 0, 0.14 and 0. | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual value was -0.62. | -0.76 (0.17)
  Change at Week 2 | -0.72 (0.23) | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual values were 0, -0.08, -3.4, -0.45, -2.37, -0.4, 0, 0 and 0. | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual value was -1.2. | -1.38 (0.23)
  Change at Week 4 | -1.03 (0.29) | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual values were -0.14, -0.51, -2, -0.74, -4.08, -1.4, 0, -0.71 and -1.14. | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual value was -0.91. | -1.77 (0.31)
  Change at Week 6: number analyzed (Participants) | 73 | 8 | 1 | 72
  Change at Week 6 | -1.17 (0.33) | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual values were -2, -0.94, -0.88, -2.94, -1.97, -3, -1 and -2. | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual value was -0.62. | -2.04 (0.34)
  Change at Week 12 | -1.51 (0.37) | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual values were -3.76, -1.8, -2.5, 0.9, -2.22, -2.4, -1.75, -0.5 and -2.75. | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual value was -2.2. | -2.10 (0.37)
  Change at Week 16: number analyzed (Participants) | 73 | 7 | 0 | 72
  Change at Week 16 | -1.37 (0.40) | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual values were -4, -2.3, -1.3, -1.9, -1, -1.33 and -3. |  | -1.92 (0.42)
  Change at Week 24: number analyzed (Participants) | 73 | 6 | 0 | 72
  Change at Week 24 | -1.04 (0.44) | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual values were -4, -1.8, -2.55, -1.15, -3 and -3. |  | -1.62 (0.43)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 20 mg; Change at Week 1: ANCOVA model for imputed datasets included treatment, region, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness) as fixed effects, and baseline average pain intensity at the index bone metastasis cancer pain site and baseline opioid dose as covariates; Test type: Superiority; p = 0.0497, ANCOVA; Difference in LS mean = -0.36, 95% CI 2-sided [-0.72 to -0.00], Standard Error of Mean 0.18
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 20 mg; Change at Week 2: ANCOVA model for imputed datasets included treatment, region, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness) as fixed effects, and baseline average pain intensity at the index bone metastasis cancer pain site and baseline opioid dose as covariates; Test type: Superiority; p = 0.0092, ANCOVA; Difference in LS mean = -0.66, 95% CI 2-sided [-1.16 to -0.17], Standard Error of Mean 0.25
Statistical Analysis 3: Comparison: Placebo vs Tanezumab 20 mg; Change at Week 4: ANCOVA model for imputed datasets included treatment, region, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness) as fixed effects, and baseline average pain intensity at the index bone metastasis cancer pain site and baseline opioid dose as covariates; Test type: Superiority; p = 0.0218, ANCOVA; Difference in LS mean = -0.74, 95% CI 2-sided [-1.37 to -0.11], Standard Error of Mean 0.32
Statistical Analysis 4: Comparison: Placebo vs Tanezumab 20 mg; Change at Week 6: ANCOVA model for imputed datasets included treatment, region, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness) as fixed effects, and baseline average pain intensity at the index bone metastasis cancer pain site and baseline opioid dose as covariates; Test type: Superiority; p = 0.0154, ANCOVA; Difference in LS mean = -0.87, 95% CI 2-sided [-1.58 to -0.17], Standard Error of Mean 0.36
Statistical Analysis 5: Comparison: Placebo vs Tanezumab 20 mg; Change at Week 12: ANCOVA model for imputed datasets included treatment, region, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness) as fixed effects, and baseline average pain intensity at the index bone metastasis cancer pain site and baseline opioid dose as covariates; Test type: Superiority; p = 0.1289, ANCOVA; Difference in LS mean = -0.59, 95% CI 2-sided [-1.36 to 0.17], Standard Error of Mean 0.39
Statistical Analysis 6: Comparison: Placebo vs Tanezumab 20 mg; Change at Week 16: ANCOVA model for imputed datasets included treatment, region, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness) as fixed effects, and baseline average pain intensity at the index bone metastasis cancer pain site and baseline opioid dose as covariates; Test type: Superiority; p = 0.2110, ANCOVA; Difference in LS mean = -0.55, 95% CI 2-sided [-1.43 to 0.32], Standard Error of Mean 0.44
Statistical Analysis 7: Comparison: Placebo vs Tanezumab 20 mg; Change at Week 24: ANCOVA model for imputed datasets included treatment, region, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness) as fixed effects, and baseline average pain intensity at the index bone metastasis cancer pain site and baseline opioid dose as covariates; Test type: Superiority; p = 0.2049, ANCOVA; Difference in LS mean = -0.58, 95% CI 2-sided [-1.49 to 0.32], Standard Error of Mean 0.46

3. Secondary Outcome: Change From Baseline in the Daily Worst Pain Intensity NRS Score in the Index Bone Metastasis Cancer Pain Site at Weeks 1, 2, 4, 6, 8, 12, 16 and 24
Description: Daily worst pain intensity in the index bone metastasis cancer pain site is assessed by participants on an 11 point pain intensity NRS ranging from 0 (no pain) to 10 (worst possible pain), higher scores signified more severity of pain. The participants describe their daily worst pain at the painful site during the past 24 hours by choosing the appropriate number from 0 to 10 on IRT diaries. Baseline daily worst pain intensity was mean of daily worst pain intensity NRS score during the baseline assessment period prior to randomization. Baseline assessment period was up to 5 days prior to dosing. The Weeks 1, 2, 4, 6, 8, 12, 16 and 24 daily worst pain intensity value was the mean of the daily worst pain intensity NRS scores recorded for each of the 7 days prior to the each specified week.
Time Frame: Baseline, Weeks 1, 2, 4, 6, 8, 12, 16 and 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Tanezumab 10 mg | Tanezumab 10/20 mg | Tanezumab 20 mg
Number analyzed (Participants) | 73 | 9 | 1 | 72
Units on a scale
  Change at Week 1 | -0.52 (0.18) | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual values were 0.4, 0.2, -2.85, -0.4, -1.8, -0.4, 0, 0.45 and 0. | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual value was -1.42. | -0.84 (0.19)
  Change at Week 2 | -0.74 (0.25) | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual values were 0.4, -0.08, -4, -0.25, -2.37, -0.4, 0, 0.6 and 0. | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual value was -1.57 | -1.47 (0.25)
  Change at Week 4 | -1.14 (0.30) | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual values were -0.02, -0.51, -1.85, -0.4, -4.08, -1.4, 0, 0.02 and -1.14. | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual value was -1.42. | -1.88 (0.31)
  Change at Week 6: number analyzed (Participants) | 73 | 8 | 1 | 72
  Change at Week 6 | -1.20 (0.33) | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual values were -2.74, -0.94, -0.54, -2.94, -1.97, -3, -0.4 and -2. | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual value was -1.14. | -2.08 (0.34)
  Change at Week 8: number analyzed (Participants) | 73 | 8 | 1 | 72
  Change at Week 8 | -1.38 (0.36) | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual values were -4.6, -1.51, -0.4, -3.65, -2.4, -3, -0.25 and -2. | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual value was -0.85. | -2.14 (0.37)
  Change at Week 12 | -1.53 (0.36) | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual values were -4.63, -1.8, -3.5, 0.6, -2.22, -2.4, -1.75, 0.1 and -2.75. | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual value was -2. | -2.25 (0.38)
  Change at Week 16: number analyzed (Participants) | 73 | 7 | 0 | 72
  Change at Week 16 | -1.32 (0.44) | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual values were -4.6, -2.3, -1.3, -1.9, -1, -0.73 and -3. |  | -2.06 (0.43)
  Change at Week 24: number analyzed (Participants) | 73 | 6 | 0 | 72
  Change at Week 24 | -1.10 (0.44) | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual values were -4.93, -1.8, -2.55, -1.15, -5.4 and -3. |  | -1.90 (0.45)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 20 mg; Change at Week 1: ANCOVA model for imputed datasets included treatment, region, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness) as fixed effects, and baseline average pain intensity at the index bone metastasis cancer pain site, baseline worst pain intensity at the index bone metastasis cancer pain site and baseline opioid dose as covariates; Test type: Superiority; p = 0.1103, ANCOVA; Difference in LS mean = -0.33, 95% CI 2-sided [-0.73 to 0.07], Standard Error of Mean 0.20
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 20 mg; Change at Week 2: ANCOVA model for imputed datasets included treatment, region, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness) as fixed effects, and baseline average pain intensity at the index bone metastasis cancer pain site, baseline worst pain intensity at the index bone metastasis cancer pain site and baseline opioid dose as covariates; Test type: Superiority; p = 0.0084, ANCOVA; Difference in LS mean = -0.73, 95% CI 2-sided [-1.26 to -0.19], Standard Error of Mean 0.27
Statistical Analysis 3: Comparison: Placebo vs Tanezumab 20 mg; Change at Week 4:ANCOVA model for imputed datasets included treatment, region, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness) as fixed effects, and baseline average pain intensity at the index bone metastasis cancer pain site, baseline worst pain intensity at the index bone metastasis cancer pain site and baseline opioid dose as covariates; Test type: Superiority; p = 0.0236, ANCOVA; Difference in LS mean = -0.75, 95% CI 2-sided [-1.39 to -0.10], Standard Error of Mean 0.33
Statistical Analysis 4: Comparison: Placebo vs Tanezumab 20 mg; Change at Week 6: ANCOVA model for imputed datasets included treatment, region, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness) as fixed effects, and baseline average pain intensity at the index bone metastasis cancer pain site, baseline worst pain intensity at the index bone metastasis cancer pain site and baseline opioid dose as covariates; Test type: Superiority; p = 0.0155, ANCOVA; Difference in LS mean = -0.88, 95% CI 2-sided [-1.59 to -0.17], Standard Error of Mean 0.36
Statistical Analysis 5: Comparison: Placebo vs Tanezumab 20 mg; Change at Week 8: ANCOVA model for imputed datasets included treatment, region, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness) as fixed effects, and baseline average pain intensity at the index bone metastasis cancer pain site, baseline worst pain intensity at the index bone metastasis cancer pain site and baseline opioid dose as covariates; Test type: Superiority; p = 0.0505, ANCOVA; Difference in LS mean = -0.76, 95% CI 2-sided [-1.52 to 0.00], Standard Error of Mean 0.38
Statistical Analysis 6: Comparison: Placebo vs Tanezumab 20 mg; Change at Week 12: ANCOVA model for imputed datasets included treatment, region, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness) as fixed effects, and baseline average pain intensity at the index bone metastasis cancer pain site, baseline worst pain intensity at the index bone metastasis cancer pain site and baseline opioid dose as covariates; Test type: Superiority; p = 0.0761, ANCOVA; Difference in LS mean = -0.72, 95% CI 2-sided [-1.52 to 0.08], Standard Error of Mean 0.40
Statistical Analysis 7: Comparison: Placebo vs Tanezumab 20 mg; Change at Week 16: ANCOVA model for imputed datasets included treatment, region, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness) as fixed effects, and baseline average pain intensity at the index bone metastasis cancer pain site, baseline worst pain intensity at the index bone metastasis cancer pain site and baseline opioid dose as covariates; Test type: Superiority; p = 0.1263, ANCOVA; Difference in LS mean = -0.74, 95% CI 2-sided [-1.70 to 0.21], Standard Error of Mean 0.48
Statistical Analysis 8: Comparison: Placebo vs Tanezumab 20 mg; Change at Week 24: ANCOVA model for imputed datasets included treatment, region, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness) as fixed effects, and baseline average pain intensity at the index bone metastasis cancer pain site, baseline worst pain intensity at the index bone metastasis cancer pain site and baseline opioid dose as covariates; Test type: Superiority; p = 0.1051, ANCOVA; Difference in LS mean = -0.79, 95% CI 2-sided [-1.76 to 0.17], Standard Error of Mean 0.49

4. Secondary Outcome: Change From Baseline in the Weekly Average Pain Intensity NRS Score in Non-Index Cancer Pain Sites at Weeks 1, 2, 4, 6, 8, 12, 16 and 24
Description: Weekly average pain intensity in the non-index cancer pain site was assessed by participants on an 11 point pain intensity NRS ranging from 0 (no pain) to 10 (worst possible pain), where higher scores signified more severity of pain. Non-index cancer pan sites were the most painful cancer pain sites other than the index bone metastasis cancer pain site. The participants described their weekly pain at the painful site by choosing the appropriate number from 0 to 10 on IRT diaries. Baseline weekly average pain intensity was weekly average pain intensity NRS score recorded on any day during the baseline assessment period. Five days prior to dosing was considered as baseline assessment period. The Weeks 1, 2, 4, 6, 8, 12, 16 and 24 weekly average pain intensity value was the weekly average pain intensity NRS scores recorded on any day from the span of 7 days prior to specified week.
Time Frame: Baseline, Weeks 1, 2, 4, 6, 8, 12, 16 and 24
Population: The mITT analysis set: participants randomized to tanezumab 20 mg or placebo SC, received at least 1dose of SC study medication. Multiple imputation method was applied. As planned summarized efficacy data for tanezumab 10 mg and 10/20 mg arms not reported; for these 2 arms individual values are reported. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure and ''number analyzed'' signifies participants evaluable at specified time points.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Tanezumab 10 mg | Tanezumab 10/20 mg | Tanezumab 20 mg
Number analyzed (Participants) | 23 | 2 | 1 | 32
Units on a scale
  Change at Week 1: number analyzed (Participants) | 23 | 1 | 1 | 32
  Change at Week 1 | -0.64 (0.42) | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual value was 1. | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual value was 0. | -1.14 (0.35)
  Change at Week 2: number analyzed (Participants) | 23 | 1 | 1 | 32
  Change at Week 2 | -0.96 (0.54) | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual value was 0.5 | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual value was 1.5 | -1.81 (0.47)
  Change at Week 4 | -1.42 (0.59) | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual value were -1 and 0. | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual value was 0.5 | -2.22 (0.52)
  Change at Week 6 | -1.76 (0.65) | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual value were -1 and -3. | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual value was 0. | -2.24 (0.56)
  Change at Week 8 | -1.79 (0.70) | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual values were -2 and -3. | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual value was -2. | -2.34 (0.62)
  Change at Week 12 | -1.64 (0.59) | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual values were -2 and -1.375. | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual values was -1. | -2.14 (0.53)
  Change at Week 16: number analyzed (Participants) | 23 | 2 | 0 | 32
  Change at Week 16 | -1.06 (0.71) | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual values were -2 and -1.375. |  | -2.27 (0.60)
  Change at Week 24: number analyzed (Participants) | 23 | 1 | 0 | 32
  Change at Week 24 | -0.87 (0.68) | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual values were -2. |  | -1.92 (0.59)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 20 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.3003, ANCOVA; Difference in LS mean = -0.50, 95% CI 2-sided [-1.47 to 0.47], Standard Error of Mean 0.48
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 20 mg; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.1603, ANCOVA; Difference in LS mean = -0.84, 95% CI 2-sided [-2.03 to 0.35], Standard Error of Mean 0.59
Statistical Analysis 3: Comparison: Placebo vs Tanezumab 20 mg; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; p = 0.2298, ANCOVA; Difference in LS mean = -0.80, 95% CI 2-sided [-2.13 to 0.53], Standard Error of Mean 0.66
Statistical Analysis 4: Comparison: Placebo vs Tanezumab 20 mg; [analysis description as in outcome 2, analysis 4]; Test type: Superiority; p = 0.5054, ANCOVA; Difference in LS mean = -0.48, 95% CI 2-sided [-1.93 to 0.97], Standard Error of Mean 0.72
Statistical Analysis 5: Comparison: Placebo vs Tanezumab 20 mg; Change at Week 8: ANCOVA model for imputed datasets included treatment, region, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness) as fixed effects, and baseline average pain intensity at the index bone metastasis cancer pain site and baseline opioid dose as covariates; Test type: Superiority; p = 0.4793, ANCOVA; Difference in LS mean = -0.55, 95% CI 2-sided [-2.10 to 1.01], Standard Error of Mean -0.77
Statistical Analysis 6: Comparison: Placebo vs Tanezumab 20 mg; [analysis description as in outcome 2, analysis 5]; Test type: Superiority; p = 0.4496, ANCOVA; Difference in LS mean = -0.50, 95% CI 2-sided [-1.83 to 0.83], Standard Error of Mean 0.66
Statistical Analysis 7: Comparison: Placebo vs Tanezumab 20 mg; [analysis description as in outcome 2, analysis 6]; Test type: Superiority; p = 0.1263, ANCOVA; Difference in least square LS mean = -1.21, 95% CI 2-sided [-2.77 to 0.36], Standard Error of Mean 0.77
Statistical Analysis 8: Comparison: Placebo vs Tanezumab 20 mg; [analysis description as in outcome 2, analysis 7]; Test type: Superiority; p = 0.1620, ANCOVA; Difference in LS mean = -1.05, 95% CI 2-sided [-2.54 to 0.44], Standard Error of Mean 0.73

5. Secondary Outcome: Change From Baseline in the Weekly Worst Pain Intensity NRS Score in Non-Index Cancer Pain Sites at Weeks 1, 2, 4, 6, 8, 12, 16 and 24
Description: Weekly worst pain intensity in the non-index cancer pain site was assessed by participants on an 11 point pain intensity NRS ranging from 0 (no pain) to 10 (worst possible pain), higher scores signified more severity of pain. Non-index cancer pan sites were the most painful cancer pain sites other than the index bone metastasis cancer pain site. The participants describe their weekly worst pain at the painful site by choosing the appropriate number from 0 to 10 on IRT diaries. Baseline weekly worst pain intensity was weekly worst pain intensity NRS score recorded on any day during the baseline assessment period. Five days prior to dosing was considered as baseline assessment period. The Weeks 1, 2, 4, 6, 8, 12, 16 and 24 weekly worst pain intensity value was the weekly worst pain intensity NRS scores which was recorded on any day from the span of 7 days prior to specified week.
Time Frame: Baseline, Weeks 1, 2, 4, 6, 8, 12, 16 and 24
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Tanezumab 10 mg | Tanezumab 10/20 mg | Tanezumab 20 mg
Number analyzed (Participants) | 23 | 2 | 1 | 32
Units on a scale
  Change at Week 1: number analyzed (Participants) | 23 | 1 | 1 | 32
  Change at Week 1 | -0.43 (0.50) | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual values was 1. | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual values was -0.5 | -1.50 (0.42)
  Change at Week 2: number analyzed (Participants) | 23 | 1 | 1 | 32
  Change at Week 2 | -0.34 (0.59) | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual values were 0.5 | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual values was 0.5. | -2.30 (0.51)
  Change at Week 4 | -1.18 (0.66) | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual values were -1 and 0. | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual values was 0. | -2.62 (0.56)
  Change at Week 6 | -1.62 (0.73) | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual values were -1 and -3. | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual values was 0.5. | -2.50 (0.61)
  Change at Week 8 | -1.77 (0.74) | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual values were -2 and -3. | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual values was -1. | -2.54 (0.64)
  Change at Week 12 | -1.36 (0.68) | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual values were -2 and -1.75. | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual values was -0.5 | -2.56 (0.57)
  Change at Week 16: number analyzed (Participants) | 23 | 2 | 0 | 32
  Change at Week 16 | -0.85 (0.82) | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual values were -2 and -1.625 |  | -2.75 (0.66)
  Change at Week 24: number analyzed (Participants) | 23 | 1 | 0 | 32
  Change at Week 24 | -0.73 (0.79) | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual value was -2. |  | -2.35 (0.67)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 20 mg; Change at Week 1: ANCOVA model for imputed datasets included treatment, region, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness) as fixed effects, and baseline average pain intensity at the index bone metastasis cancer pain site, baseline worst pain intensity at the non-index cancer pain sites and baseline opioid dose as covariates; Test type: Superiority; p = 0.0575, ANCOVA; Difference in LS mean = -1.07, 95% CI 2-sided [-2.17 to 0.04], Standard Error of Mean 0.54
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 20 mg; Change at Week 2: ANCOVA model for imputed datasets included treatment, region, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness) as fixed effects, and baseline average pain intensity at the index bone metastasis cancer pain site, baseline worst pain intensity at the non-index cancer pain sites and baseline opioid dose as covariates; Test type: Superiority; p = 0.0031, ANCOVA; Difference in LS mean = -1.96, 95% CI 2-sided [-3.22 to -0.70], Standard Error of Mean 0.62
Statistical Analysis 3: Comparison: Placebo vs Tanezumab 20 mg; Change at Week 4: ANCOVA model for imputed datasets included treatment, region, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness) as fixed effects, and baseline average pain intensity at the index bone metastasis cancer pain site, baseline worst pain intensity at the non-index cancer pain sites and baseline opioid dose as covariates; Test type: Superiority; p = 0.0410, ANCOVA; Difference in LS mean = -1.44, 95% CI 2-sided [-2.82 to -0.06], Standard Error of Mean 0.68
Statistical Analysis 4: Comparison: Placebo vs Tanezumab 20 mg; Change at Week 6: ANCOVA model for imputed datasets included treatment, region, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness) as fixed effects, and baseline average pain intensity at the index bone metastasis cancer pain site, baseline worst pain intensity at the non-index cancer pain sites and baseline opioid dose as covariates; Test type: Superiority; p = 0.2598, ANCOVA; Difference in LS mean = -0.88, 95% CI 2-sided [-2.44 to 0.68], Standard Error of Mean 0.77
Statistical Analysis 5: Comparison: Placebo vs Tanezumab 20 mg; Change at Week 8: ANCOVA model for imputed datasets included treatment, region, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness) as fixed effects, and baseline average pain intensity at the index bone metastasis cancer pain site, baseline worst pain intensity at the non-index cancer pain sites and baseline opioid dose as covariates; Test type: Superiority; p = 0.3426, ANCOVA; Difference in LS mean = -0.77, 95% CI 2-sided [-2.38 to 0.85], Standard Error of Mean 0.80
Statistical Analysis 6: Comparison: Placebo vs Tanezumab 20 mg; Change at Week 12: ANCOVA model for imputed datasets included treatment, region, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness) as fixed effects, and baseline average pain intensity at the index bone metastasis cancer pain site, baseline worst pain intensity at the non-index cancer pain sites and baseline opioid dose as covariates; Test type: Superiority; p = 0.1034, ANCOVA; Difference in LS mean = -1.20, 95% CI 2-sided [-2.65 to 0.26], Standard Error of Mean 0.72
Statistical Analysis 7: Comparison: Placebo vs Tanezumab 20 mg; Change at Week 16: ANCOVA model for imputed datasets included treatment, region, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness) as fixed effects, and baseline average pain intensity at the index bone metastasis cancer pain site, baseline worst pain intensity at the non-index cancer pain sites and baseline opioid dose as covariates; Test type: Superiority; p = 0.0290, ANCOVA; Difference in LS mean = -1.91, 95% CI 2-sided [-3.60 to -0.21], Standard Error of Mean 0.84
Statistical Analysis 8: Comparison: Placebo vs Tanezumab 20 mg; Change at Week 24: ANCOVA model for imputed datasets included treatment, region, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness) as fixed effects, and baseline average pain intensity at the index bone metastasis cancer pain site, baseline worst pain intensity at the non-index cancer pain sites and baseline opioid dose as covariates; Test type: Superiority; p = 0.0600, ANCOVA; Difference in LS mean = -1.62, 95% CI 2-sided [-3.31 to 0.07], Standard Error of Mean 0.83

6. Secondary Outcome: Change From Baseline in the Daily Average Pain Intensity NRS Score in the Non-Index Visceral Cancer Pain Sites at Weeks 1, 2, 4, 6, 8, 12, 16 and 24
Description: Daily average pain intensity in the non-index visceral cancer pain site was assessed by participants on an 11 point pain intensity NRS ranging from 0 (no pain) to 10 (worst possible pain), where higher scores signified more severity of pain. The participants described their pain at the painful site during the past 24 hours by choosing the appropriate number from 0 to 10 on IRT diaries. Baseline is defined as the mean average daily pain intensity NRS score during the baseline assessment period prior to randomization. The Weeks 1, 2, 4, 6, 8, 12, 16 and 24 pain intensity value is the mean of the daily average pain intensity scores for the 7 days prior to the each specified week.
Time Frame: Baseline, Weeks 1, 2, 4, 6, 8, 12, 16 and 24
Population: Participant with non-index visceral cancer pain sites were less than 10, hence data was not collected and analysis was not performed for this outcome measure.
Arm/Group | Placebo | Tanezumab 20 mg | Tanezumab 10 mg | Tanezumab 10/20 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Secondary Outcome: Change From Baseline in the Daily Worst Pain Intensity NRS Score in the Non-Index Visceral Cancer Pain Sites at Weeks 1, 2, 4, 6, 8, 12, 16 and 24
Description: Daily worst pain intensity in the index bone metastasis cancer pain site was assessed by participants on an 11 point pain intensity NRS ranging from 0 (no pain) to 10 (worst possible pain), where higher scores signified more severity of pain. The participants recorded their daily worst pain at the painful site during the past 24 hours by choosing the appropriate number from 0 to 10 on IRT diaries. Baseline pain intensity value was mean of the daily worst pain intensity NRS scores during the baseline assessment period prior to randomization. Baseline assessment period was up to 5 days prior to dosing. The Weeks 1, 2, 4, 6, 8, 12, 16 and 24 pain intensity value is the mean of the daily worst pain intensity scores for the 7 days prior to the each specified week.
Time Frame: Baseline, Weeks 1, 2, 4, 6, 8, 12, 16 and 24
Population: as for outcome 6
Arm/Group | Placebo | Tanezumab 10 mg | Tanezumab 10/20 mg | Tanezumab 20 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With Cumulative Reduction of >=30, 50, 70 and 90 Percent (%) From Baseline in Daily Average Pain Intensity NRS Score in the Index Bone Metastasis Cancer Pain Site at Weeks 1, 2, 4, 6, 8, 12, 16 and 24
Description: Daily average pain intensity in the index bone metastasis cancer pain site was assessed by participants on an 11 point pain intensity NRS ranging from 0 (no pain) to 10 (worst possible pain), where higher scores = more severity of pain. The participants recorded their daily average pain at the painful site during the past 24 hours by choosing the appropriate number from 0 to 10 on IRT diaries. The Weeks 1, 2, 4, 6, 8, 12, 16 and 24 pain intensity value = mean of the daily average pain intensity NRS scores for the 7 days prior to the each week. Number of participants with cumulative reduction of >= 30, 50, 70, and 90 % in daily average pain intensity NRS score in the index bone metastasis cancer pain site from Baseline to Weeks 1, 2, 4, 6, 8, 12, 16 and 24 were reported. Participants might be reported more than once in the specified rows for a time point. Rows with only non-zero data for cumulative reduction at specified time points, for at least 1 reporting arm, are reported below.
Time Frame: Baseline, Weeks 1, 2, 4, 6, 8, 12, 16 and 24
Population: The mITT analysis set was analyzed. Mixed Baseline Observation Carried Forward (BOCF)/ Last Observation Carried Forward (LOCF) imputation was applied. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure and ''number analyzed'' signifies participants evaluable at specified time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 10 mg | Tanezumab 10/20 mg | Tanezumab 20 mg
Number analyzed (Participants) | 73 | 9 | 1 | 71
Participants
  Week 1: Reduction of >=30% | 8 | 2 | 0 | 9
  Week 1: Reduction of >=50% | 4 | 0 | 0 | 4
  Week 1: Reduction of >=70% | 0 | 0 | 0 | 1
  Week 2: Reduction of >=30% | 11 | 2 | 0 | 18
  Week 2: Reduction of >=50% | 3 | 1 | 0 | 13
  Week 2: Reduction of >=70% | 0 | 0 | 0 | 4
  Week 2: Reduction of >=90% | 0 | 0 | 0 | 2
  Week 4: Reduction of >=30% | 18 | 2 | 0 | 25
  Week 4: Reduction of >=50% | 6 | 1 | 0 | 16
  Week 4: Reduction of >=70% | 2 | 1 | 0 | 9
  Week 4: Reduction of >=90% | 0 | 0 | 0 | 3
  Week 6: Reduction of >=30%: number analyzed (Participants) | 73 | 8 | 1 | 71
  Week 6: Reduction of >=30% | 20 | 5 | 0 | 30
  Week 6: Reduction of >=50%: number analyzed (Participants) | 73 | 8 | 1 | 71
  Week 6: Reduction of >=50% | 6 | 1 | 0 | 19
  Week 6: Reduction of >=70%: number analyzed (Participants) | 73 | 8 | 1 | 71
  Week 6: Reduction of >=70% | 2 | 0 | 0 | 10
  Week 6: Reduction of >=90%: number analyzed (Participants) | 73 | 8 | 1 | 71
  Week 6: Reduction of >=90% | 0 | 0 | 0 | 3
  Week 8: Reduction of >=30%: number analyzed (Participants) | 73 | 8 | 1 | 71
  Week 8: Reduction of >=30% | 19 | 5 | 0 | 28
  Week 8: Reduction of >=50%: number analyzed (Participants) | 73 | 8 | 1 | 71
  Week 8: Reduction of >=50% | 9 | 2 | 0 | 18
  Week 8: Reduction of >=70%: number analyzed (Participants) | 73 | 8 | 1 | 71
  Week 8: Reduction of >=70% | 3 | 0 | 0 | 9
  Week 8: Reduction of >=90%: number analyzed (Participants) | 73 | 8 | 1 | 71
  Week 8: Reduction of >=90% | 1 | 0 | 0 | 5
  Week 12: Reduction of >=30% | 21 | 5 | 1 | 32
  Week 12: Reduction of >=50% | 12 | 2 | 0 | 21
  Week 12: Reduction of >=70% | 6 | 1 | 0 | 10
  Week 12: Reduction of >=90% | 2 | 0 | 0 | 5
  Week 16: Reduction of >=30%: number analyzed (Participants) | 73 | 7 | 0 | 71
  Week 16: Reduction of >=30% | 17 | 2 |  | 27
  Week 16: Reduction of >=50%: number analyzed (Participants) | 73 | 7 | 0 | 71
  Week 16: Reduction of >=50% | 12 | 2 |  | 19
  Week 16: Reduction of >=70%: number analyzed (Participants) | 73 | 7 | 0 | 71
  Week 16: Reduction of >=70% | 7 | 1 |  | 12
  Week 16: Reduction of >=90%: number analyzed (Participants) | 73 | 7 | 0 | 71
  Week 16: Reduction of >=90% | 5 | 0 |  | 5
  Week 24: Reduction of >=30%: number analyzed (Participants) | 73 | 6 | 0 | 71
  Week 24: Reduction of >=30% | 16 | 4 |  | 27
  Week 24: Reduction of >=50%: number analyzed (Participants) | 73 | 6 | 0 | 71
  Week 24: Reduction of >=50% | 10 | 3 |  | 19
  Week 24: Reduction of >=70%: number analyzed (Participants) | 73 | 6 | 0 | 71
  Week 24: Reduction of >=70% | 5 | 1 |  | 11
  Week 24: Reduction of >=90%: number analyzed (Participants) | 73 | 6 | 0 | 71
  Week 24: Reduction of >=90% | 3 | 0 |  | 4
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 20 mg; Week 1 Reduction >=30%: Logistic regression model included baseline average pain intensity at the index bone metastasis cancer pain site, treatment, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness); Test type: Superiority; p = 0.8054, Regression, Logistic; Odds Ratio (OR) = 1.14, 95% CI 2-sided [0.41 to 3.18]
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 20 mg; Week 1 Reduction >=50%: Logistic regression model included baseline average pain intensity at the index bone metastasis cancer pain site, treatment, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness); Test type: Superiority; p = 0.9292, Regression, Logistic; Odds Ratio (OR) = 0.94, 95% CI 2-sided [0.22 to 3.98]
Statistical Analysis 3: Comparison: Placebo vs Tanezumab 20 mg; Week 1 Reduction >=70%: Logistic regression model included baseline average pain intensity at the index bone metastasis cancer pain site, treatment, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness); Test type: Superiority; p = 0.9565, Regression, Logistic
Statistical Analysis 4: Comparison: Placebo vs Tanezumab 20 mg; Week 2 Reduction >=30%: Logistic regression model included baseline average pain intensity at the index bone metastasis cancer pain site, treatment, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness); Test type: Superiority; p = 0.1429, Regression, Logistic; Odds Ratio (OR) = 1.88, 95% CI 2-sided [0.81 to 4.36]
Statistical Analysis 5: Comparison: Placebo vs Tanezumab 20 mg; Week 2 Reduction >=50%: Logistic regression model included baseline average pain intensity at the index bone metastasis cancer pain site, treatment, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness); Test type: Superiority; p = 0.0140, Regression, Logistic; Odds Ratio (OR) = 5.19, 95% CI [1.40 to 19.31]
Statistical Analysis 6: Comparison: Placebo vs Tanezumab 20 mg; Week 2 Reduction >=70%: Logistic regression model included baseline average pain intensity at the index bone metastasis cancer pain site, treatment, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness); Test type: Superiority; p = 0.9450, Regression, Logistic
Statistical Analysis 7: Comparison: Placebo vs Tanezumab 20 mg; Week 2 Reduction >=90%: Logistic regression model included baseline average pain intensity at the index bone metastasis cancer pain site, treatment, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness); Test type: Superiority; p = 0.9489, Regression, Logistic
Statistical Analysis 8: Comparison: Placebo vs Tanezumab 20 mg; Week 4 Reduction >=30%: Logistic regression model included baseline average pain intensity at the index bone metastasis cancer pain site, treatment, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness); Test type: Superiority; p = 0.1932, Regression, Logistic; Odds Ratio (OR) = 1.63, 95% CI 2-sided [0.78 to 3.39]
Statistical Analysis 9: Comparison: Placebo vs Tanezumab 20 mg; Week 4 Reduction >=50%: Logistic regression model included baseline average pain intensity at the index bone metastasis cancer pain site, treatment, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness); Test type: Superiority; p = 0.0254, Regression, Logistic; Odds Ratio (OR) = 3.17, 95% CI 2-sided [1.15 to 8.74]
Statistical Analysis 10: Comparison: Placebo vs Tanezumab 20 mg; Week 4 Reduction >=70%: Logistic regression model included baseline average pain intensity at the index bone metastasis cancer pain site, treatment, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness); Test type: Superiority; p = 0.0455, Regression, Logistic; Odds Ratio (OR) = 5.00, 95% CI 2-sided [1.03 to 24.16]
Statistical Analysis 11: Comparison: Placebo vs Tanezumab 20 mg; Week 4 Reduction >=90%: Logistic regression model included baseline average pain intensity at the index bone metastasis cancer pain site, treatment, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness); Test type: Superiority; p = 0.9464, Regression, Logistic
Statistical Analysis 12: Comparison: Placebo vs Tanezumab 20 mg; Week 6 Reduction >=30%: Logistic regression model included baseline average pain intensity at the index bone metastasis cancer pain site, treatment, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness); Test type: Superiority; p = 0.0969, Regression, Logistic; Odds Ratio (OR) = 1.83, 95% CI 2-sided [0.90 to 3.72]
Statistical Analysis 13: Comparison: Placebo vs Tanezumab 20 mg; Week 6 Reduction >=50%: Logistic regression model included baseline average pain intensity at the index bone metastasis cancer pain site, treatment, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness); Test type: Superiority; p = 0.0043, Regression, Logistic; Odds Ratio (OR) = 4.31, 95% CI 2-sided [1.58 to 11.74]
Statistical Analysis 14: Comparison: Placebo vs Tanezumab 20 mg; Week 6 Reduction >=70%: Logistic regression model included baseline average pain intensity at the index bone metastasis cancer pain site, treatment, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness); Test type: Superiority; p = 0.0352, Regression, Logistic; Odds Ratio (OR) = 5.49, 95% CI 2-sided [1.13 to 26.75]
Statistical Analysis 15: Comparison: Placebo vs Tanezumab 20 mg; Week 6 Reduction >=90%: Logistic regression model included baseline average pain intensity at the index bone metastasis cancer pain site, treatment, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness); Test type: Superiority; p = 0.9464, Regression, Logistic
Statistical Analysis 16: Comparison: Placebo vs Tanezumab 20 mg; Week 8 Reduction >=30%: Logistic regression model included baseline average pain intensity at the index bone metastasis cancer pain site, treatment, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness); Test type: Superiority; p = 0.1471, Regression, Logistic; Odds Ratio (OR) = 1.71, 95% CI 2-sided [0.83 to 3.52]
Statistical Analysis 17: Comparison: Placebo vs Tanezumab 20 mg; Week 8 Reduction >=50%: Logistic regression model included baseline average pain intensity at the index bone metastasis cancer pain site, treatment, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness); Test type: Superiority; p = 0.0405, Regression, Logistic; Odds Ratio (OR) = 2.55, 95% CI 2-sided [1.04 to 6.22]
Statistical Analysis 18: Comparison: Placebo vs Tanezumab 20 mg; Week 8 Reduction >=70%: Logistic regression model included baseline average pain intensity at the index bone metastasis cancer pain site, treatment, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness); Test type: Superiority; p = 0.0993, Regression, Logistic; Odds Ratio (OR) = 3.21, 95% CI 2-sided [0.80 to 12.83]
Statistical Analysis 19: Comparison: Placebo vs Tanezumab 20 mg; Week 8 Reduction >=90%: Logistic regression model included baseline average pain intensity at the index bone metastasis cancer pain site, treatment, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness); Test type: Superiority; p = 0.1726, Regression, Logistic; Odds Ratio (OR) = 4.71, 95% CI 2-sided [0.51 to 43.64]
Statistical Analysis 20: Comparison: Placebo vs Tanezumab 20 mg; Week 12 Reduction >=30%: Logistic regression model included baseline average pain intensity at the index bone metastasis cancer pain site, treatment, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness); Test type: Superiority; p = 0.0918, Regression, Logistic; Odds Ratio (OR) = 1.84, 95% CI 2-sided [0.91 to 3.74]
Statistical Analysis 21: Comparison: Placebo vs Tanezumab 20 mg; Week 12 Reduction >=50%: Logistic regression model included baseline average pain intensity at the index bone metastasis cancer pain site, treatment, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness); Test type: Superiority; p = 0.0704, Regression, Logistic; Odds Ratio (OR) = 2.13, 95% CI 2-sided [0.94 to 4.82]
Statistical Analysis 22: Comparison: Placebo vs Tanezumab 20 mg; Week 12 Reduction >=70%: Logistic regression model included baseline average pain intensity at the index bone metastasis cancer pain site, treatment, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness); Test type: Superiority; p = 0.3569, Regression, Logistic; Odds Ratio (OR) = 1.67, 95% CI 2-sided [0.56 to 5.01]
Statistical Analysis 23: Comparison: Placebo vs Tanezumab 20 mg; Week 12 Reduction >=90%: Logistic regression model included baseline average pain intensity at the index bone metastasis cancer pain site, treatment, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness); Test type: Superiority; p = 0.3062, Regression, Logistic; Odds Ratio (OR) = 2.46, 95% CI 2-sided [0.44 to 13.79]
Statistical Analysis 24: Comparison: Placebo vs Tanezumab 20 mg; Week 16 Reduction >=30%: Logistic regression model included baseline average pain intensity at the index bone metastasis cancer pain site, treatment, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness); Test type: Superiority; p = 0.1058, Regression, Logistic; Odds Ratio (OR) = 1.84, 95% CI 2-sided [0.88 to 3.85]
Statistical Analysis 25: Comparison: Placebo vs Tanezumab 20 mg; Week 16 Reduction >=50%: Logistic regression model included baseline average pain intensity at the index bone metastasis cancer pain site, treatment, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness); Test type: Superiority; p = 0.1571, Regression, Logistic; Odds Ratio (OR) = 1.81, 95% CI 2-sided [0.79 to 4.14]
Statistical Analysis 26: Comparison: Placebo vs Tanezumab 20 mg; Week 16 Reduction >=70%: Logistic regression model included baseline average pain intensity at the index bone metastasis cancer pain site, treatment, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness); Test type: Superiority; p = 0.2454, Regression, Logistic; Odds Ratio (OR) = 1.85, 95% CI 2-sided [0.65 to 5.24]
Statistical Analysis 27: Comparison: Placebo vs Tanezumab 20 mg; Week 16 Reduction >=90%: Logistic regression model included baseline average pain intensity at the index bone metastasis cancer pain site, treatment, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness); Test type: Superiority; p = 0.8867, Regression, Logistic; Odds Ratio (OR) = 0.91, 95% CI 2-sided [0.24 to 3.46]
Statistical Analysis 28: Comparison: Placebo vs Tanezumab 20 mg; Week 24 Reduction >=30%: Logistic regression model included baseline average pain intensity at the index bone metastasis cancer pain site, treatment, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness); Test type: Superiority; p = 0.0689, Regression, Logistic; Odds Ratio (OR) = 2.00, 95% CI 2-sided [0.95 to 4.21]
Statistical Analysis 29: Comparison: Placebo vs Tanezumab 20 mg; Week 24 Reduction >=50%: Logistic regression model included baseline average pain intensity at the index bone metastasis cancer pain site, treatment, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness); Test type: Superiority; p = 0.0568, Regression, Logistic; Odds Ratio (OR) = 2.30, 95% CI 2-sided [0.98 to 5.44]
Statistical Analysis 30: Comparison: Placebo vs Tanezumab 20 mg; Week 24 Reduction >=70%: Logistic regression model included baseline average pain intensity at the index bone metastasis cancer pain site, treatment, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness); Test type: Superiority; p = 0.1268, Regression, Logistic; Odds Ratio (OR) = 2.41, 95% CI 2-sided [0.78 to 7.46]
Statistical Analysis 31: Comparison: Placebo vs Tanezumab 20 mg; Week 24 Reduction >=90%: Logistic regression model included baseline average pain intensity at the index bone metastasis cancer pain site, treatment, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness); Test type: Superiority; p = 0.7971, Regression, Logistic; Odds Ratio (OR) = 1.23, 95% CI 2-sided [0.25 to 6.00]

9. Secondary Outcome: Number of Participants With Reduction of >=30, 50, 70 and 90% From Baseline in Daily Worst Pain Intensity NRS Score in the Index Bone Metastasis Cancer Pain Site at Weeks 1, 2, 4, 6, 8, 12, 16 and 24
Description: Daily worst pain intensity in the index bone metastasis cancer pain site was assessed by participants on an 11 point pain intensity NRS ranging from 0 (no pain) to 10 (worst possible pain), where higher scores = more severity of pain. The participants recorded their daily worst pain at the painful site during the past 24 hours by choosing the appropriate number from 0 to 10 on IRT diaries. The Weeks 1, 2, 4, 6, 8, 12, 16 and 24 pain intensity value = mean of the daily worst pain intensity NRS scores for the 7 days prior to the each week. Number of participants with cumulative reduction of >= 30, 50, 70, and 90 % in daily worst pain intensity NRS score in the index bone metastasis cancer pain site from Baseline to Weeks 1, 2, 4, 6, 8, 12, 16 and 24 were reported. Participants might be reported more than once in the specified rows for a time point. Rows with only non-zero data for cumulative reduction at specified time points, for at least 1 reporting arm, are reported below.
Time Frame: Baseline, Weeks 1, 2, 4, 6, 8, 12, 16 and 24
Population: The mITT analysis set was analyzed. Multiple imputation method was applied. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure and ''number analyzed'' signifies participants evaluable at specified time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 10 mg | Tanezumab 10/20 mg | Tanezumab 20 mg
Number analyzed (Participants) | 73 | 9 | 1 | 71
Participants
  Week 1: Reduction of >=30% | 7 | 2 | 0 | 9
  Week 1: Reduction of >=50% | 1 | 0 | 0 | 3
  Week 1: Reduction of >=70% | 0 | 0 | 0 | 2
  Week 1: Reduction of >=90% | 0 | 0 | 0 | 0
  Week 2: Reduction of >=30% | 9 | 2 | 0 | 17
  Week 2: Reduction of >=50% | 2 | 1 | 0 | 8
  Week 2: Reduction of >=70% | 0 | 0 | 0 | 5
  Week 2: Reduction of >=90% | 0 | 0 | 0 | 2
  Week 4: Reduction of >=30% | 12 | 1 | 0 | 21
  Week 4: Reduction of >=50% | 5 | 1 | 0 | 14
  Week 4: Reduction of >=70% | 0 | 1 | 0 | 6
  Week 4: Reduction of >=90% | 0 | 0 | 0 | 2
  Week 6: Reduction of >=30%: number analyzed (Participants) | 73 | 8 | 1 | 71
  Week 6: Reduction of >=30% | 13 | 4 | 0 | 26
  Week 6: Reduction of >=50%: number analyzed (Participants) | 73 | 8 | 1 | 71
  Week 6: Reduction of >=50% | 4 | 1 | 0 | 14
  Week 6: Reduction of >=70%: number analyzed (Participants) | 73 | 8 | 1 | 71
  Week 6: Reduction of >=70% | 2 | 0 | 0 | 7
  Week 6: Reduction of >=90%: number analyzed (Participants) | 73 | 8 | 1 | 71
  Week 6: Reduction of >=90% | 0 | 0 | 0 | 2
  Week 8: Reduction of >=30%: number analyzed (Participants) | 73 | 8 | 1 | 71
  Week 8: Reduction of >=30% | 14 | 5 | 0 | 24
  Week 8: Reduction of >=50%: number analyzed (Participants) | 73 | 8 | 1 | 71
  Week 8: Reduction of >=50% | 7 | 2 | 0 | 16
  Week 8: Reduction of >=70%: number analyzed (Participants) | 73 | 8 | 1 | 71
  Week 8: Reduction of >=70% | 2 | 0 | 0 | 8
  Week 8: Reduction of >=90%: number analyzed (Participants) | 73 | 8 | 1 | 71
  Week 8: Reduction of >=90% | 2 | 0 | 0 | 2
  Week 12: Reduction of >=30% | 16 | 5 | 0 | 24
  Week 12: Reduction of >=50% | 8 | 2 | 0 | 16
  Week 12: Reduction of >=70% | 5 | 1 | 0 | 7
  Week 12: Reduction of >=90% | 2 | 0 | 0 | 4
  Week 16: Reduction of >=30%: number analyzed (Participants) | 73 | 7 | 0 | 71
  Week 16: Reduction of >=30% | 11 | 2 |  | 24
  Week 16: Reduction of >=50%: number analyzed (Participants) | 73 | 7 | 0 | 71
  Week 16: Reduction of >=50% | 9 | 2 |  | 18
  Week 16: Reduction of >=70%: number analyzed (Participants) | 73 | 7 | 0 | 71
  Week 16: Reduction of >=70% | 7 | 0 |  | 11
  Week 16: Reduction of >=90%: number analyzed (Participants) | 73 | 7 | 0 | 71
  Week 16: Reduction of >=90% | 3 | 0 |  | 3
  Week 24: Reduction of >=30%: number analyzed (Participants) | 73 | 6 | 0 | 71
  Week 24: Reduction of >=30% | 11 | 4 |  | 25
  Week 24: Reduction of >=50%: number analyzed (Participants) | 73 | 6 | 0 | 71
  Week 24: Reduction of >=50% | 9 | 3 |  | 18
  Week 24: Reduction of >=70%: number analyzed (Participants) | 73 | 6 | 0 | 71
  Week 24: Reduction of >=70% | 4 | 2 |  | 9
  Week 24: Reduction of >=90%: number analyzed (Participants) | 73 | 6 | 0 | 71
  Week 24: Reduction of >=90% | 2 | 0 |  | 3
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 20 mg; Week 1 Reduction >=30%: Logistic regression model included baseline average pain intensity at the index bone metastasis cancer pain site, baseline worst pain intensity at the index bone metastasis cancer pain site, treatment, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness); Test type: Superiority; p = 0.6658, Regression, Logistic; Odds Ratio (OR) = 1.27, 95% CI 2-sided [0.43 to 3.70]
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 20 mg; Week 1 Reduction >=50%: Logistic regression model included baseline average pain intensity at the index bone metastasis cancer pain site, baseline worst pain intensity at the index bone metastasis cancer pain site, treatment, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness); Test type: Superiority; p = 0.3443, Regression, Logistic; Odds Ratio (OR) = 3.07, 95% CI 2-sided [0.30 to 31.35]
Statistical Analysis 3: Comparison: Placebo vs Tanezumab 20 mg; Week 1 Reduction >=70%: Logistic regression model included baseline average pain intensity at the index bone metastasis cancer pain site, baseline worst pain intensity at the index bone metastasis cancer pain site, treatment, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness); Test type: Superiority; p = 0.9527, Regression, Logistic
Statistical Analysis 4: Comparison: Placebo vs Tanezumab 20 mg; Week 2 Reduction >=30%: Logistic regression model included baseline average pain intensity at the index bone metastasis cancer pain site, baseline worst pain intensity at the index bone metastasis cancer pain site, treatment, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness); Test type: Superiority; p = 0.0757, Regression, Logistic; Odds Ratio (OR) = 2.25, 95% CI 2-sided [0.92 to 5.50]
Statistical Analysis 5: Comparison: Placebo vs Tanezumab 20 mg; Week 2 Reduction >=50%: Logistic regression model included baseline average pain intensity at the index bone metastasis cancer pain site, baseline worst pain intensity at the index bone metastasis cancer pain site, treatment, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness); Test type: Superiority; p = 0.0659, Regression, Logistic; Odds Ratio (OR) = 4.51, 95% CI 2-sided [0.91 to 22.42]
Statistical Analysis 6: Comparison: Placebo vs Tanezumab 20 mg; Week 2 Reduction >=70%: Logistic regression model included baseline average pain intensity at the index bone metastasis cancer pain site, baseline worst pain intensity at the index bone metastasis cancer pain site, treatment, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness); Test type: Superiority; p = 0.9380, Regression, Logistic
Statistical Analysis 7: Comparison: Placebo vs Tanezumab 20 mg; Week 2 Reduction >=90%: Logistic regression model included baseline average pain intensity at the index bone metastasis cancer pain site, baseline worst pain intensity at the index bone metastasis cancer pain site, treatment, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness); Test type: Superiority; p = 0.9493, Regression, Logistic
Statistical Analysis 8: Comparison: Placebo vs Tanezumab 20 mg; Week 4 Reduction >=30%: Logistic regression model included baseline average pain intensity at the index bone metastasis cancer pain site, baseline worst pain intensity at the index bone metastasis cancer pain site, treatment, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness); Test type: Superiority; p = 0.0914, Regression, Logistic; Odds Ratio (OR) = 2.02, 95% CI 2-sided [0.89 to 4.59]
Statistical Analysis 9: Comparison: Placebo vs Tanezumab 20 mg; Week 4 Reduction >=50%: Logistic regression model included baseline average pain intensity at the index bone metastasis cancer pain site, baseline worst pain intensity at the index bone metastasis cancer pain site, treatment, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness); Test type: Superiority; p = 0.0359, Regression, Logistic; Odds Ratio (OR) = 3.22, 95% CI 2-sided [1.08 to 9.61]
Statistical Analysis 10: Comparison: Placebo vs Tanezumab 20 mg; Week 4 Reduction >=70%: Logistic regression model included baseline average pain intensity at the index bone metastasis cancer pain site, baseline worst pain intensity at the index bone metastasis cancer pain site, treatment, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness); Test type: Superiority; p = 0.9538, Regression, Logistic
Statistical Analysis 11: Comparison: Placebo vs Tanezumab 20 mg; Week 4 Reduction >=90%: Logistic regression model included baseline average pain intensity at the index bone metastasis cancer pain site, baseline worst pain intensity at the index bone metastasis cancer pain site, treatment, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness); Test type: Superiority; p = 0.9493, Regression, Logistic
Statistical Analysis 12: Comparison: Placebo vs Tanezumab 20 mg; Week 6 Reduction >=30%: Logistic regression model included baseline average pain intensity at the index bone metastasis cancer pain site, baseline worst pain intensity at the index bone metastasis cancer pain site, treatment, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness); Test type: Superiority; p = 0.0143, Regression, Logistic; Odds Ratio (OR) = 2.66, 95% CI 2-sided [1.22 to 5.80]
Statistical Analysis 13: Comparison: Placebo vs Tanezumab 20 mg; Week 6 Reduction >=50%: Logistic regression model included baseline average pain intensity at the index bone metastasis cancer pain site, baseline worst pain intensity at the index bone metastasis cancer pain site, treatment, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness); Test type: Superiority; p = 0.0176, Regression, Logistic; Odds Ratio (OR) = 4.20, 95% CI 2-sided [1.28 to 13.74]
Statistical Analysis 14: Comparison: Placebo vs Tanezumab 20 mg; Week 6 Reduction >=70%: Logistic regression model included baseline average pain intensity at the index bone metastasis cancer pain site, baseline worst pain intensity at the index bone metastasis cancer pain site, treatment, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness); Test type: Superiority; p = 0.1298, Regression, Logistic; Odds Ratio (OR) = 3.53, 95% CI 2-sided [0.69 to 18.06]
Statistical Analysis 15: Comparison: Placebo vs Tanezumab 20 mg; Week 6 Reduction >=90%: Logistic regression model included baseline average pain intensity at the index bone metastasis cancer pain site, baseline worst pain intensity at the index bone metastasis cancer pain site, treatment, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness); Test type: Superiority; p = 0.9493, Regression, Logistic
Statistical Analysis 16: Comparison: Placebo vs Tanezumab 20 mg; Week 8 Reduction >=30%: Logistic regression model included baseline average pain intensity at the index bone metastasis cancer pain site, baseline worst pain intensity at the index bone metastasis cancer pain site, treatment, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness); Test type: Superiority; p = 0.0527, Regression, Logistic; Odds Ratio (OR) = 2.15, 95% CI 2-sided [0.99 to 4.67]
Statistical Analysis 17: Comparison: Placebo vs Tanezumab 20 mg; Week 8 Reduction >=50%: Logistic regression model included baseline average pain intensity at the index bone metastasis cancer pain site, baseline worst pain intensity at the index bone metastasis cancer pain site, treatment, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness); Test type: Superiority; p = 0.0457, Regression, Logistic; Odds Ratio (OR) = 2.69, 95% CI 2-sided [1.02 to 7.12]
Statistical Analysis 18: Comparison: Placebo vs Tanezumab 20 mg; Week 8 Reduction >=70%: Logistic regression model included baseline average pain intensity at the index bone metastasis cancer pain site, baseline worst pain intensity at the index bone metastasis cancer pain site, treatment, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness); Test type: Superiority; p = 0.0994, Regression, Logistic; Odds Ratio (OR) = 3.91, 95% CI 2-sided [0.77 to 19.76]
Statistical Analysis 19: Comparison: Placebo vs Tanezumab 20 mg; Week 8 Reduction >=90%: Logistic regression model included baseline average pain intensity at the index bone metastasis cancer pain site, baseline worst pain intensity at the index bone metastasis cancer pain site, treatment, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness); Test type: Superiority; p = 0.6977, Regression, Logistic; Odds Ratio (OR) = 0.65, 95% CI 2-sided [0.07 to 5.86]
Statistical Analysis 20: Comparison: Placebo vs Tanezumab 20 mg; Week 12 Reduction >=30%: Logistic regression model included baseline average pain intensity at the index bone metastasis cancer pain site, baseline worst pain intensity at the index bone metastasis cancer pain site, treatment, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness); Test type: Superiority; p = 0.1460, Regression, Logistic; Odds Ratio (OR) = 1.76, 95% CI 2-sided [0.82 to 3.75]
Statistical Analysis 21: Comparison: Placebo vs Tanezumab 20 mg; Week 12 Reduction >=50%: Logistic regression model included baseline average pain intensity at the index bone metastasis cancer pain site, baseline worst pain intensity at the index bone metastasis cancer pain site, treatment, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness); Test type: Superiority; p = 0.0742, Regression, Logistic; Odds Ratio (OR) = 2.35, 95% CI 2-sided [0.92 to 6.01]
Statistical Analysis 22: Comparison: Placebo vs Tanezumab 20 mg; Week 12 Reduction >=70%: Logistic regression model included baseline average pain intensity at the index bone metastasis cancer pain site, baseline worst pain intensity at the index bone metastasis cancer pain site, treatment, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness); Test type: Superiority; p = 0.5565, Regression, Logistic; Odds Ratio (OR) = 1.44, 95% CI 2-sided [0.42 to 4.91]
Statistical Analysis 23: Comparison: Placebo vs Tanezumab 20 mg; Week 12 Reduction >=90%: Logistic regression model included baseline average pain intensity at the index bone metastasis cancer pain site, baseline worst pain intensity at the index bone metastasis cancer pain site, treatment, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness); Test type: Superiority; p = 0.5623, Regression, Logistic; Odds Ratio (OR) = 1.70, 95% CI 2-sided [0.28 to 10.35]
Statistical Analysis 24: Comparison: Placebo vs Tanezumab 20 mg; Week 16 Reduction >=30%: Logistic regression model included baseline average pain intensity at the index bone metastasis cancer pain site, baseline worst pain intensity at the index bone metastasis cancer pain site, treatment, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness); Test type: Superiority; p = 0.0116, Regression, Logistic; Odds Ratio (OR) = 2.86, 95% CI 2-sided [1.27 to 6.47]
Statistical Analysis 25: Comparison: Placebo vs Tanezumab 20 mg; Week 16 Reduction >=50%: Logistic regression model included baseline average pain intensity at the index bone metastasis cancer pain site, baseline worst pain intensity at the index bone metastasis cancer pain site, treatment, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness); Test type: Superiority; p = 0.0615, Regression, Logistic; Odds Ratio (OR) = 2.34, 95% CI 2-sided [0.96 to 5.70]
Statistical Analysis 26: Comparison: Placebo vs Tanezumab 20 mg; Week 16 Reduction >=70%: Logistic regression model included baseline average pain intensity at the index bone metastasis cancer pain site, baseline worst pain intensity at the index bone metastasis cancer pain site, treatment, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness); Test type: Superiority; p = 0.3316, Regression, Logistic; Odds Ratio (OR) = 1.68, 95% CI 2-sided [0.59 to 4.80]
Statistical Analysis 27: Comparison: Placebo vs Tanezumab 20 mg; Week 16 Reduction >=90%: Logistic regression model included baseline average pain intensity at the index bone metastasis cancer pain site, baseline worst pain intensity at the index bone metastasis cancer pain site, treatment, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness); Test type: Superiority; p = 0.9946, Regression, Logistic; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.19 to 5.33]
Statistical Analysis 28: Comparison: Placebo vs Tanezumab 20 mg; Week 24 Reduction >=30%: Logistic regression model included baseline average pain intensity at the index bone metastasis cancer pain site, baseline worst pain intensity at the index bone metastasis cancer pain site, treatment, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness); Test type: Superiority; p = 0.0083, Regression, Logistic; Odds Ratio (OR) = 2.99, 95% CI 2-sided [1.33 to 6.76]
Statistical Analysis 29: Comparison: Placebo vs Tanezumab 20 mg; Week 24 Reduction >=50%: Logistic regression model included baseline average pain intensity at the index bone metastasis cancer pain site, baseline worst pain intensity at the index bone metastasis cancer pain site, treatment, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness); Test type: Superiority; p = 0.0513, Regression, Logistic; Odds Ratio (OR) = 2.42, 95% CI 2-sided [1.00 to 5.88]
Statistical Analysis 30: Comparison: Placebo vs Tanezumab 20 mg; Week 24 Reduction >=70%: Logistic regression model included baseline average pain intensity at the index bone metastasis cancer pain site, baseline worst pain intensity at the index bone metastasis cancer pain site, treatment, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness); Test type: Superiority; p = 0.1528, Regression, Logistic; Odds Ratio (OR) = 2.48, 95% CI 2-sided [0.71 to 8.58]
Statistical Analysis 31: Comparison: Placebo vs Tanezumab 20 mg; Week 24 Reduction >=90%: Logistic regression model included baseline average pain intensity at the index bone metastasis cancer pain site, baseline worst pain intensity at the index bone metastasis cancer pain site, treatment, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness); Test type: Superiority; p = 0.7251, Regression, Logistic; Odds Ratio (OR) = 1.41, 95% CI 2-sided [0.21 to 9.65]

10. Secondary Outcome: Change From Baseline in Participant's Global Assessment of Cancer Pain (PGA-CP) at Weeks 2, 4, 8, 16 and 24
Description: Participants at specified time points, answered to the following question, "Considering all the ways your cancer pain affects you, how are you doing today?" on a Likert scale ranging from 1 to 5, on IRT diaries. Scores: 1= very good (asymptomatic and no limitation of normal activities); 2= good (mild symptoms and no limitation of normal activities); 3= fair (moderate symptoms and limitation of some normal activities); 4= poor (severe symptoms and inability to carry out most normal activities); and 5= very poor (very severe symptoms which are intolerable and inability to carry out all normal activities). Higher scores signified worsening of condition.
Time Frame: Baseline, Weeks 2, 4, 8, 16 and 24
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Groups:
- Tanezumab 10mg: Participants in this discontinued treatment arm, received tanezumab 10 mg SC once every 8 weeks before protocol amendment 3 and completed their treatment before the amendment.
Arm/Group | Placebo | Tanezumab 10mg | Tanezumab 10/20 mg | Tanezumab 20 mg
Number analyzed (Participants) | 73 | 9 | 1 | 71
Units on a scale
  Change at Week 2 | -0.39 (0.11) | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual values were 0, 0, -3, 0, -2, 1, 0, -1 and -1. | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual values was 1. | -0.43 (0.12)
  Change at Week 4 | -0.36 (0.14) | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual values were 0, 1, 0, 0, -3, 1, 0, 0 and -1. | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual values was 0. | -0.66 (0.14)
  Change at Week 8 | -0.23 (0.16) | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual values were -1, 0, -1, 0, -3, 1, 0, -1 and -1. | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual values was 1. | -0.56 (0.17)
  Change at Week 16: number analyzed (Participants) | 73 | 6 | 0 | 71
  Change at Week 16 | -0.16 (0.16) | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual values were -2, 0, -3, 1, 0 and -1. |  | -0.32 (0.17)
  Change at Week 24: number analyzed (Participants) | 73 | 6 | 0 | 71
  Change at Week 24 | -0.19 (0.18) | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual values were -1, 0, -3, 1, 2 and -1. |  | -0.29 (0.17)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 20 mg; Change at Week 2: ANCOVA model for imputed datasets included treatment, region, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness) as fixed effects, and baseline global assessment score, baseline average pain intensity at the index bone metastasis cancer pain site, and baseline opioid dose as covariates; Test type: Superiority; p = 0.7045, ANCOVA; Difference in LS mean = -0.04, 95% CI 2-sided [-0.28 to 0.19], Standard Error of Mean 0.12
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 20 mg; Change at Week 4: ANCOVA model for imputed datasets included treatment, region, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness) as fixed effects, and baseline global assessment score, baseline average pain intensity at the index bone metastasis cancer pain site, and baseline opioid dose as covariates; Test type: Superiority; p = 0.0402, ANCOVA; Difference in LS mean = -0.30, 95% CI 2-sided [-0.59 to -0.01], Standard Error of Mean 0.14
Statistical Analysis 3: Comparison: Placebo vs Tanezumab 20 mg; Change at Week 8: ANCOVA model for imputed datasets included treatment, region, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness) as fixed effects, and baseline global assessment score, baseline average pain intensity at the index bone metastasis cancer pain site, and baseline opioid dose as covariates; Test type: Superiority; p = 0.0637, ANCOVA; Difference in LS mean = -0.33, 95% CI 2-sided [-0.67 to 0.02], Standard Error of Mean 0.17
Statistical Analysis 4: Comparison: Placebo vs Tanezumab 20 mg; Change at Week 16: ANCOVA model for imputed datasets included treatment, region, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness) as fixed effects, and baseline global assessment score, baseline average pain intensity at the index bone metastasis cancer pain site, and baseline opioid dose as covariates; Test type: Superiority; p = 0.3804, ANCOVA; Difference in LS mean = -0.16, 95% CI 2-sided [-0.53 to 0.20], Standard Error of Mean 0.18
Statistical Analysis 5: Comparison: Placebo vs Tanezumab 20 mg; Change at Week 24: ANCOVA model for imputed datasets included treatment, region, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness) as fixed effects, and baseline global assessment score, baseline average pain intensity at the index bone metastasis cancer pain site, and baseline opioid dose as covariates; Test type: Superiority; p = 0.5894, ANCOVA; Difference in LS mean = -0.10, 95% CI 2-sided [-0.47 to 0.27], Standard Error of Mean 0.18

11. Secondary Outcome: Number of Participants With Reduction of >=2 Points From Baseline in PGA-CP Scores at Weeks 2, 4, 8, 16 and 24
Description: Participants at specified time points, answered to the following question, "Considering all the ways your cancer pain affects you, how are you doing today?" on a Likert scale ranging from 1 to 5, on IRT diaries. Scores:1= very good (asymptomatic and no limitation of normal activities); 2= good (mild symptoms and no limitation of normal activities); 3= fair (moderate symptoms and limitation of some normal activities); 4= poor (severe symptoms and inability to carry out most normal activities); and 5= very poor (very severe symptoms which are intolerable and inability to carry out all normal activities). Higher scores signified worsening of condition.
Time Frame: Baseline, Weeks 2, 4, 8, 16 and 24
Population: The mITT analysis set: participants randomized to tanezumab 20 mg or placebo SC, received at least 1dose of SC study medication. Multiple imputation method was applied. Here, ''number analyzed'' signifies participants evaluable at specified time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 10 mg | Tanezumab 10/20 mg | Tanezumab 20 mg
Number analyzed (Participants) | 73 | 9 | 1 | 72
Participants
  Week 2 | 7 | 2 | 0 | 5
  Week 4 | 9 | 1 | 0 | 11
  Week 8 | 10 | 1 | 0 | 12
  Week 16: number analyzed (Participants) | 73 | 6 | 0 | 72
  Week 16 | 9 | 2 |  | 12
  Week 24: number analyzed (Participants) | 73 | 6 | 0 | 72
  Week 24 | 9 | 1 |  | 11
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 20 mg; Week 2: Logistic regression model included baseline PGA-CP, baseline average pain intensity at the index bone metastasis cancer pain site, treatment, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness); Test type: Superiority; p = 0.2033, Regression, Logistic; Odds Ratio (OR) = 0.38, 95% CI 2-sided [0.09 to 1.69]
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 20 mg; Week 4: Logistic regression model included baseline PGA-CP, baseline average pain intensity at the index bone metastasis cancer pain site, treatment, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness); Test type: Superiority; p = 0.7627, Regression, Logistic; Odds Ratio (OR) = 1.18, 95% CI 2-sided [0.41 to 3.41]
Statistical Analysis 3: Comparison: Placebo vs Tanezumab 20 mg; Week 8: Logistic regression model included baseline PGA-CP, baseline average pain intensity at the index bone metastasis cancer pain site, treatment, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness); Test type: Superiority; p = 0.6894, Regression, Logistic; Odds Ratio (OR) = 1.23, 95% CI 2-sided [0.44 to 3.43]
Statistical Analysis 4: Comparison: Placebo vs Tanezumab 20 mg; Week 16: Logistic regression model included baseline PGA-CP, baseline average pain intensity at the index bone metastasis cancer pain site, treatment, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness); Test type: Superiority; p = 0.5905, Regression, Logistic; Odds Ratio (OR) = 1.34, 95% CI 2-sided [0.47 to 3.83]
Statistical Analysis 5: Comparison: Placebo vs Tanezumab 20 mg; Week 24: Logistic regression model included baseline PGA-CP, baseline average pain intensity at the index bone metastasis cancer pain site, treatment, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness); Test type: Superiority; p = 0.8354, Regression, Logistic; Odds Ratio (OR) = 1.12, 95% CI 2-sided [0.38 to 3.35]

12. Secondary Outcome: Average Daily Total Opioid Consumption at Weeks 1, 2, 4, 6, 8, 12, 16 and 24
Description: In this outcome measure average daily opioid consumption was reported in milligram of morphine equivalent dose (mg of MED).
Time Frame: Weeks 1, 2, 4, 6, 8, 12, 16 and 24
Population: The mITT analysis set: participants randomized to tanezumab 20 mg or placebo SC, received at least 1dose of SC study medication. LOCF data was applied. As planned summarized efficacy data for tanezumab 10 mg and 10/20 mg arms not reported; for these 2 arms individual values are reported. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure and ''number analyzed'' signifies participants evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: mg of MED
Arm/Group | Placebo | Tanezumab 10 mg | Tanezumab 10/20 mg | Tanezumab 20 mg
Number analyzed (Participants) | 73 | 9 | 1 | 72
mg of MED
  Week 1: number analyzed (Participants) | 72 | 9 | 1 | 69
  Week 1 | 183.94 (275.05) | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as Mean and SD. Individual values were 0.3, 30, 181.54, 1082.74, 122.03, 10, 120, 22.5 and 30. | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as Mean and SD. Individual values was 510. | 186.86 (351.83)
  Week 2: number analyzed (Participants) | 73 | 9 | 1 | 69
  Week 2 | 177.98 (270.67) | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as Mean and SD. Individual values were 0.3, 30, 182.4, 1082.22, 120.96, 10, 120, 22.5 and 30. | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as Mean and SD. Individual values was 510. | 188.41 (356.15)
  Week 4: number analyzed (Participants) | 73 | 9 | 1 | 69
  Week 4 | 177.87 (266.93) | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as Mean and SD. Individual values were 0.3, 34.28, 182.4, 1082.22, 120.96, 52.85, 120, 22.5 and 30. | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as Mean and SD. Individual values was 480. | 181.32 (349.82)
  Week 6: number analyzed (Participants) | 73 | 9 | 1 | 70
  Week 6 | 186.20 (280.44) | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as Mean and SD. Individual values were 0.3, 95, 182.4, 1081.54, 120.96, 10, 137.14, 22.5 and 30. | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as Mean and SD. Individual values was 510. | 173.45 (346.27)
  Week 8: number analyzed (Participants) | 73 | 9 | 1 | 70
  Week 8 | 188.10 (281.01) | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as Mean and SD. Individual values were 0.3, 122.14, 2.4, 1081.71, 120.96, 10, 120, 22.5 and 30. | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as Mean and SD. Individual values was 510. | 170.31 (327.19)
  Week 12: number analyzed (Participants) | 73 | 9 | 1 | 70
  Week 12 | 187.43 (336.74) | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as Mean and SD. Individual values were 0.3, 258.57, 2.4, 1.2, 88.45, 10, 120, 22.5 and 30. | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as Mean and SD. Individual values was 480. | 177.06 (332.39)
  Week 16: number analyzed (Participants) | 73 | 9 | 1 | 70
  Week 16 | 189.62 (333.77) | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as Mean and SD. Individual values were 0.3, 170, 2.4, 1.2, 86.31, 10, 120, 22.5 and 30. | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as Mean and SD. Individual values was 480. | 173.48 (329.17)
  Week 24: number analyzed (Participants) | 73 | 9 | 1 | 70
  Week 24 | 189.78 (353.10) | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as Mean and SD. Individual values were 0.3, 170, 2.4, 1.2, 88.45, 74.28, 120, 18.21 and 30. | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as Mean and SD. Individual values was 480. | 346.95 (1537.00)

13. Secondary Outcome: Average Number of Doses of Rescue Opioid Consumption at Weeks 1, 2, 4, 6, 8, 12, 16 and 24
Description: In this outcome measure average number of doses of rescue opioid consumption at specified time points were reported.
Time Frame: Weeks 1, 2, 4, 6, 8, 12, 16 and 24
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Doses
Arm/Group | Placebo | Tanezumab 10 mg | Tanezumab 10/20 mg | Tanezumab 20 mg
Number analyzed (Participants) | 73 | 9 | 1 | 72
Doses
  Week 1: number analyzed (Participants) | 52 | 8 | 1 | 42
  Week 1 | 1.15 (0.76) | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as Mean and SD. Individual values were 1, 1, 1, 1, 0.14, 1,1 and 1. | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as Mean and SD. Individual values was 1. | 0.96 (0.48)
  Week 2: number analyzed (Participants) | 54 | 8 | 1 | 44
  Week 2 | 1.11 (0.69) | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as Mean and SD. Individual values were 1, 1, 1, 1, 0.14, 1,1 and 1. | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as Mean and SD. Individual values was 1. | 0.89 (0.52)
  Week 4: number analyzed (Participants) | 56 | 9 | 1 | 46
  Week 4 | 1.08 (0.69) | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as Mean and SD. Individual values were 1, 1, 1, 1, 0.14, 0.14, 0.85,1 and 1. | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as Mean and SD. Individual values was 0.43. | 0.80 (0.57)
  Week 6: number analyzed (Participants) | 61 | 9 | 1 | 48
  Week 6 | 0.95 (0.70) | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as Mean and SD. Individual values were 1, 1, 1, 0.85, 0.14, 0.14, 1, 1 and 1. | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as Mean and SD. Individual values was 1. | 0.80 (0.65)
  Week 8: number analyzed (Participants) | 61 | 9 | 1 | 48
  Week 8 | 0.99 (0.72) | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as Mean and SD. Individual values were 1, 1, 1, 1, 0.28, 0.14, 0.71, 1 and 1. | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as Mean and SD. Individual values was 1. | 0.81 (0.61)
  Week 12: number analyzed (Participants) | 61 | 9 | 1 | 48
  Week 12 | 0.92 (0.94) | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as Mean and SD. Individual values were 1, 1, 1, 1, 1, 0.14, 0.14, 1 and 1. | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as Mean and SD. Individual values was 1. | 0.73 (0.57)
  Week 16: number analyzed (Participants) | 62 | 9 | 1 | 48
  Week 16 | 0.86 (0.93) | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as Mean and SD. Individual values were 1, 1, 1, 1, 0.85, 0.14, 0.14, 1 and 1. | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as Mean and SD. Individual values was 1. | 0.75 (0.57)
  Week 24: number analyzed (Participants) | 65 | 9 | 1 | 49
  Week 24 | 0.79 (0.93) | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as Mean and SD. Individual values were 1, 1, 1, 1, 1, 0.14, 0.14, 0.42 and 1. | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as Mean and SD. Individual values was 1. | 0.69 (0.57)

14. Secondary Outcome: Change From Baseline in the Weekly Opioid-Related Symptom Distress Scale (OR-SDS) at Weeks 2, 4, 8, 16, and 24
Description: OR-SDS: questionnaire evaluated opioid-related 12 symptoms. For each symptom, participants assigned integer scores to assess severity (none =0 to very severe =4), distress (none =0 to very much =5), and frequency (none =0 to almost constantly =4; participants reported number of retching/vomiting episodes (none =0, 1-2 episodes =1, 3-4 episodes =2, 5-6 episodes =3, >6 episodes =4). Frequency composite score: mean of frequency scores from all symptoms, ranged from 0 (none) to 4 (almost constantly); higher scores = worse condition. Severity composite score: mean of severity scores from all 12 symptoms, ranged from 0 (none) to 4 (maximum severity); higher scores = worse condition. Distress composite score: mean of distress scores from all 12 symptoms, ranged from 0 (none) to 5 (maximum distress); higher scores = worse condition. Multi domain average (MDA): average of each symptom for frequency, severity, and distress; ranged from 0 (none) to 4.34 (worse); higher scores = worse condition.
Time Frame: Baseline, Weeks 2, 4, 8, 16, and 24
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Tanezumab 10mg | Tanezumab 10/20 mg | Tanezumab 20 mg
Number analyzed (Participants) | 73 | 2 | 1 | 72
Units on a scale
  Change at Week 2: Frequency Composite Score | -0.06 (0.16) | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual values were -1 and -0.6. | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual values was -1.33. | -0.11 (0.17)
  Change at Week 2: Severity Composite Score | -0.18 (0.11) | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual values were 0 and 0.2. | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual values was -0.83. | -0.02 (0.12)
  Change at Week 2: Distress Composite Score | -0.08 (0.18) | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual values were -1 and -0.25. | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual values was 0.17. | 0.09 (0.19)
  Change at Week 2: MDA Composite Score | -0.10 (0.14) | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual values were -0.67 and -0.22. | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual values was -0.67. | -0.02 (0.15)
  Change at Week 4: Frequency Composite Score: number analyzed (Participants) | 73 | 1 | 1 | 72
  Change at Week 4: Frequency Composite Score | -0.19 (0.14) | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual values were -0.8. | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual values was -1.5. | -0.12 (0.14)
  Change at Week 4: Severity Composite Score: number analyzed (Participants) | 73 | 1 | 1 | 72
  Change at Week 4: Severity Composite Score | -0.10 (0.12) | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual values were 0. | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual values was -0.5. | -0.01 (0.13)
  Change at Week 4: Distress Composite Score: number analyzed (Participants) | 73 | 1 | 1 | 72
  Change at Week 4: Distress Composite Score | 0.12 (0.15) | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual values were -0.25. | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual values was 0. | 0.11 (0.15)
  Change at Week 4: MDA Composite Score: number analyzed (Participants) | 73 | 1 | 1 | 72
  Change at Week 4: MDA Composite Score | -0.06 (0.12) | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual values were -0.35. | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual values was -0.67. | -0.00 (0.13)
  Change at Week 8: Frequency Composite Score | 0.07 (0.15) | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual values were -1 and 0. | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual values was -1. | -0.10 (0.16)
  Change at Week 8: Severity Composite Score | -0.07 (0.12) | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual values were 0 and 0. | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual values was -0.75. | -0.17 (0.13)
  Change at Week 8: Distress Composite Score | 0.03 (0.19) | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual values were -1 and -0.25. | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual values was 0.25. | 0.26 (0.20)
  Change at Week 8: MDA Composite Score | 0.02 (0.13) | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual values were -0.67 and -0.08. | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual values was -0.5. | -0.02 (0.14)
  Change at Week 16: Frequency Composite Score: number analyzed (Participants) | 73 | 1 | 0 | 72
  Change at Week 16: Frequency Composite Score | 0.08 (0.19) | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual values were -1. |  | -0.07 (0.22)
  Change at Week 16: Severity Composite Score: number analyzed (Participants) | 73 | 1 | 0 | 72
  Change at Week 16: Severity Composite Score | -0.12 (0.15) | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual values were 0. |  | 0.08 (0.17)
  Change at Week 16: Distress Composite Score: number analyzed (Participants) | 73 | 1 | 0 | 72
  Change at Week 16: Distress Composite Score | 0.10 (0.20) | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual values were -0.75. |  | -0.07 (0.24)
  Change at Week 16: MDA Composite Score: number analyzed (Participants) | 73 | 1 | 0 | 72
  Change at Week 16: MDA Composite Score | 0.02 (0.16) | NA (NA) — Data for this arm was not summarized per plan. Hence, not reported as LS mean and SE. Individual values were -0.58. |  | -0.04 (0.19)
  Change at Week 24: Frequency Composite Score: number analyzed (Participants) | 73 | 0 | 0 | 72
  Change at Week 24: Frequency Composite Score | 0.29 (0.21) |  |  | -0.13 (0.24)
  Change at Week 24: Severity Composite Score: number analyzed (Participants) | 73 | 0 | 0 | 72
  Change at Week 24: Severity Composite Score | -0.01 (0.17) |  |  | 0.16 (0.18)
  Change at Week 24: Distress Composite Score: number analyzed (Participants) | 73 | 0 | 0 | 72
  Change at Week 24: Distress Composite Score | 0.33 (0.21) |  |  | 0.22 (0.23)
  Change at Week 24: MDA Composite Score: number analyzed (Participants) | 73 | 0 | 0 | 72
  Change at Week 24: MDA Composite Score | 0.17 (0.18) |  |  | 0.07 (0.20)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 20 mg; Week 2 Frequency Composite Score: Mixed model for repeated measurements (MMRM) model includes time (study week), treatment, region, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness) as fixed effects, and treatment*time interaction, baseline OR-SDS frequency scores, and baseline average pain intensity at the index bone metastasis cancer pain site as covariates; Test type: Superiority; p = 0.8069, Mixed Models Analysis; Difference in LS mean = -0.05, 95% CI 2-sided [-0.49 to 0.38], Standard Error of Mean 0.22
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 20 mg; Week 4 Frequency Composite Score: MMRM model includes time (study week), treatment, region, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness) as fixed effects, and treatment*time interaction, baseline OR-SDS frequency scores, and baseline average pain intensity at the index bone metastasis cancer pain site as covariates; Test type: Superiority; p = 0.7127, Mixed Models Analysis; Difference in LS mean = 0.06, 95% CI 2-sided [-0.28 to 0.41], Standard Error of Mean 0.17
Statistical Analysis 3: Comparison: Placebo vs Tanezumab 20 mg; Week 8 Frequency Composite Score: MMRM model includes time (study week), treatment, region, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness) as fixed effects, and treatment*time interaction, baseline OR-SDS frequency scores, and baseline average pain intensity at the index bone metastasis cancer pain site as covariates; Test type: Superiority; p = 0.3933, Mixed Models Analysis; Difference in LS mean = -0.17, 95% CI 2-sided [-0.57 to 0.23], Standard Error of Mean 0.20
Statistical Analysis 4: Comparison: Placebo vs Tanezumab 20 mg; Week 16 Frequency Composite Score: MMRM model includes time (study week), treatment, region, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness) as fixed effects, and treatment*time interaction, baseline OR-SDS frequency scores, and baseline average pain intensity at the index bone metastasis cancer pain site as covariates; Test type: Superiority; p = 0.5869, Mixed Models Analysis; Difference in LS mean = -0.15, 95% CI 2-sided [-0.71 to 0.41], Standard Error of Mean 0.28
Statistical Analysis 5: Comparison: Placebo vs Tanezumab 20 mg; Week 24 Frequency Composite Score: MMRM model includes time (study week), treatment, region, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness) as fixed effects, and treatment*time interaction, baseline OR-SDS frequency scores, and baseline average pain intensity at the index bone metastasis cancer pain site as covariates; Test type: Superiority; p = 0.1814, Mixed Models Analysis; Difference in LS mean = -0.42, 95% CI 2-sided [-1.05 to 0.21], Standard Error of Mean 0.30
Statistical Analysis 6: Comparison: Placebo vs Tanezumab 20 mg; Week 2 Severity Composite Score: MMRM model includes time (study week), treatment, region, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness) as fixed effects, and treatment*time interaction, baseline OR-SDS severity scores, and baseline average pain intensity at the index bone metastasis cancer pain site as covariates; Test type: Superiority; p = 0.2822, Mixed Models Analysis; Difference in LS mean = 0.16, 95% CI 2-sided [-0.14 to 0.46], Standard Error of Mean 0.15
Statistical Analysis 7: Comparison: Placebo vs Tanezumab 20 mg; Week 4 Severity Composite Score: MMRM model includes time (study week), treatment, region, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness) as fixed effects, and treatment*time interaction, baseline OR-SDS severity scores, and baseline average pain intensity at the index bone metastasis cancer pain site as covariates; Test type: Superiority; p = 0.5795, Mixed Models Analysis; Difference in LS mean = 0.09, 95% CI 2-sided [-0.23 to 0.41], Standard Error of Mean 0.16
Statistical Analysis 8: Comparison: Placebo vs Tanezumab 20 mg; Week 8 Severity Composite Score: MMRM model includes time (study week), treatment, region, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness) as fixed effects, and treatment*time interaction, baseline OR-SDS severity scores, and baseline average pain intensity at the index bone metastasis cancer pain site as covariates; Test type: Superiority; p = 0.5486, Mixed Models Analysis; Difference in LS mean = -0.10, 95% CI 2-sided [-0.42 to 0.22], Standard Error of Mean 0.16
Statistical Analysis 9: Comparison: Placebo vs Tanezumab 20 mg; Week 16 Severity Composite Score: MMRM model includes time (study week), treatment, region, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness) as fixed effects, and treatment*time interaction, baseline OR-SDS severity scores, and baseline average pain intensity at the index bone metastasis cancer pain site as covariates; Test type: Superiority; p = 0.3692, Mixed Models Analysis; Difference in LS mean = 0.20, 95% CI 2-sided [-0.24 to 0.63], Standard Error of Mean 0.22
Statistical Analysis 10: Comparison: Placebo vs Tanezumab 20 mg; Week 24 Severity Composite Score: MMRM model includes time (study week), treatment, region, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness) as fixed effects, and treatment*time interaction, baseline OR-SDS severity scores, and baseline average pain intensity at the index bone metastasis cancer pain site as covariates; Test type: Superiority; p = 0.4724, Mixed Models Analysis; Difference in LS mean = 0.17, 95% CI 2-sided [-0.30 to 0.63], Standard Error of Mean 0.23
Statistical Analysis 11: Comparison: Placebo vs Tanezumab 20 mg; Week 2 Distress Composite Score: MMRM model includes time (study week), treatment, region, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness) as fixed effects, and treatment*time interaction, baseline OR-SDS distress scores, and baseline average pain intensity at the index bone metastasis cancer pain site as covariates; Test type: Superiority; p = 0.4770, Mixed Models Analysis; Difference in LS mean = 0.17, 95% CI 2-sided [-0.30 to 0.64], Standard Error of Mean 0.23
Statistical Analysis 12: Comparison: Placebo vs Tanezumab 20 mg; Week 4 Distress Composite Score: MMRM model includes time (study week), treatment, region, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness) as fixed effects, and treatment*time interaction, baseline OR-SDS distress scores, and baseline average pain intensity at the index bone metastasis cancer pain site as covariates; Test type: Superiority; p = 0.9791, Mixed Models Analysis; Difference in LS mean = -0.00, 95% CI 2-sided [-0.38 to 0.37], Standard Error of Mean 0.18
Statistical Analysis 13: Comparison: Placebo vs Tanezumab 20 mg; Week 8 Distress Composite Score: MMRM model includes time (study week), treatment, region, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness) as fixed effects, and treatment*time interaction, baseline OR-SDS distress scores, and baseline average pain intensity at the index bone metastasis cancer pain site as covariates; Test type: Superiority; p = 0.3574, Mixed Models Analysis; Difference in LS mean = 0.23, 95% CI 2-sided [-0.27 to 0.74], Standard Error of Mean 0.25
Statistical Analysis 14: Comparison: Placebo vs Tanezumab 20 mg; Week 16 Distress Composite Score: MMRM model includes time (study week), treatment, region, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness) as fixed effects, and treatment*time interaction, baseline OR-SDS distress scores, and baseline average pain intensity at the index bone metastasis cancer pain site as covariates; Test type: Superiority; p = 0.5607, Mixed Models Analysis; Difference in LS mean = 0.17, 95% CI 2-sided [-0.77 to 0.42], Standard Error of Mean 0.29
Statistical Analysis 15: Comparison: Placebo vs Tanezumab 20 mg; Week 24 Distress Composite Score: MMRM model includes time (study week), treatment, region, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness) as fixed effects, and treatment*time interaction, baseline OR-SDS distress scores, and baseline average pain intensity at the index bone metastasis cancer pain site as covariates; Test type: Superiority; p = 0.7143, Mixed Models Analysis; Difference in LS mean = -0.10, 95% CI 2-sided [-0.68 to 0.47], Standard Error of Mean 0.28
Statistical Analysis 16: Comparison: Placebo vs Tanezumab 20 mg; Week 2 MDA Composite Score: MMRM model includes time (study week), treatment, region, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness) as fixed effects, and treatment*time interaction, baseline OR-SDS MDA scores, and baseline average pain intensity at the index bone metastasis cancer pain site as covariates; Test type: Superiority; p = 0.6381, Mixed Models Analysis; Difference in LS mean = 0.09, 95% CI 2-sided [-0.28 to 0.45], Standard Error of Mean 0.18
Statistical Analysis 17: Comparison: Placebo vs Tanezumab 20 mg; Week 4 MDA Composite Score: MMRM model includes time (study week), treatment, region, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness) as fixed effects, and treatment*time interaction, baseline OR-SDS MDA scores, and baseline average pain intensity at the index bone metastasis cancer pain site as covariates; Test type: Superiority; p = 0.7181, Mixed Models Analysis; Difference in LS mean = 0.06, 95% CI 2-sided [-0.25 to 0.37], Standard Error of Mean 0.15
Statistical Analysis 18: Comparison: Placebo vs Tanezumab 20 mg; Week 8 MDA Composite Score: MMRM model includes time (study week), treatment, region, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness) as fixed effects, and treatment*time interaction, baseline OR-SDS MDA scores, and baseline average pain intensity at the index bone metastasis cancer pain site as covariates; Test type: Superiority; p = 0.8378, Mixed Models Analysis; Difference in least square (LS) mean = -0.04, 95% CI 2-sided [-0.38 to 0.31], Standard Error of Mean 0.17
Statistical Analysis 19: Comparison: Placebo vs Tanezumab 20 mg; Week 16 MDA Composite Score: MMRM model includes time (study week), treatment, region, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness) as fixed effects, and treatment*time interaction, baseline OR-SDS MDA scores, and baseline average pain intensity at the index bone metastasis cancer pain site as covariates; Test type: Superiority; p = 0.7950, Mixed Models Analysis; Difference in LS mean = -0.06, 95% CI 2-sided [-0.52 to 0.40], Standard Error of Mean 0.23
Statistical Analysis 20: Comparison: Placebo vs Tanezumab 20 mg; Week 24 MDA Composite Score: MMRM model includes time (study week), treatment, region, and randomization stratification variables (concomitant anticancer treatment and tumor aggressiveness) as fixed effects, and treatment*time interaction, baseline OR-SDS MDA scores, and baseline average pain intensity at the index bone metastasis cancer pain site as covariates; Test type: Superiority; p = 0.6719, Mixed Models Analysis; Difference in LS mean = -0.11, 95% CI 2-sided [-0.62 to 0.40], Standard Error of Mean 0.25

15. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between first dose of study drug and up to 24 weeks post last dose that were absent before treatment or that worsened relative to pretreatment state. AEs included both serious and all non-serious AEs. Participants were followed up to 24 weeks after study drug last dose.
Time Frame: Day 1 of dosing up to 24 weeks post last dose (maximum up to Week 48)
Population: The safety analysis set was defined as all participants treated with tanezumab or placebo SC, including participants who received tanezumab 10 mg prior to protocol amendment 3.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 10 mg | Tanezumab 10/20 mg | Tanezumab 20 mg
Number analyzed (Participants) | 73 | 9 | 1 | 72
Participants | 52 | 9 | 1 | 62

16. Secondary Outcome: Number of Participants With Laboratory Abnormalities (Normal Baseline)
Description: Laboratory abnormality criteria included: hemoglobin (HGB); hematocrit; erythrocytes < 0.8*lower limit of normal (LLN); erythrocyte mean corpuscular volume/HGB/ HGB concentration, erythrocytes distribution width <0.9*LLN, >1.1*upper limit of normal (ULN); platelets <0.5*LLN,>1.75* ULN; leukocytes<0.6*LLN, >1.5*ULN; lymphocytes, neutrophils <0.8*LLN, >1.2*ULN; basophils, eosinophils, monocytes >1.2*ULN; total bilirubin>1.5*ULN; activated partial thromboplastin time, prothrombin time, prothrombin intl. normalized ratio >1.1*ULN; bilirubin >1.5*ULN; aspartate aminotransferase (AT), alanine AT, gamma glutamyl transferase, lactate dehydrogenase, alkaline phosphatase >3.0*ULN; protein; albumin<0.8*LLN, >1.2*ULN; urea nitrogen, creatinine, cholesterol, triglycerides >1.3*ULN; urate >1.2*ULN; sodium <0.95*LLN,>1.05*ULN; potassium, chloride, calcium, magnesium, bicarbonate <0.9*LLN, >1.1*ULN; phosphate <0.8*LLN, >1.2*ULN; Urine: glucose, ketones, protein, HGB, bilirubin, nitrite >=1.
Time Frame: Baseline (Day 1, before dosing) up to Week 48
Population: The safety analysis set was analyzed. Here, "Overall Number of Participants Analyzed" signifies participants with a normal baseline with at least one observation of the given laboratory test while on the study. There were no participants in reporting arm "Tanezumab10/20 mg", who met the criteria for data collection and analysis of this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 10 mg | Tanezumab 10/20 mg | Tanezumab 20 mg
Number analyzed (Participants) | 42 | 8 | 0 | 50
Participants | 18 | 1 |  | 20

17. Secondary Outcome: Number of Participants With Laboratory Abnormalities (Abnormal Baseline)
Description: Laboratory abnormality criteria included: HGB; hematocrit; erythrocytes < 0.8* LLN; erythrocyte mean corpuscular volume/HGB/ HGB concentration, erythrocytes distribution width <0.9*LLN, >1.1*upper limit of normal (ULN); platelets <0.5*LLN,>1.75* ULN; leukocytes <0.6*LLN, >1.5*ULN; lymphocytes, neutrophils <0.8*LLN, >1.2*ULN; basophils, eosinophils, monocytes >1.2*ULN; activated partial thromboplastin time, prothrombin time >1.1*ULN; bilirubin>1.5*ULN; aspartate AT, alanine AT, gamma glutamyl transferase, lactate dehydrogenase, alkaline phosphatase >3.0*ULN; protein; albumin<0.8*LLN, >1.2*ULN; urea nitrogen, cholesterol, triglycerides >1.3*ULN; urate >1.2*ULN; sodium <0.95*LLN,>1.05*ULN; potassium, chloride, calcium, magnesium, bicarbonate <0.9*LLN, >1.1*ULN; phosphate <0.8*LLN, >1.2*ULN; glucose <0.6*LLN, >1.5*ULN; creatine kinase >2.0*ULN.
Time Frame: Baseline (Day 1, before dosing) up to Week 48
Population: The safety analysis set was analyzed. Here, "Overall Number of Participants Analyzed" signifies participants with an abnormal baseline with at least one observation of the given laboratory test while on the study. There were no participants in reporting arm "Tanezumab10/20 mg", who met the criteria for data collection and analysis of this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 10 mg | Tanezumab 10/20 mg | Tanezumab 20 mg
Number analyzed (Participants) | 38 | 8 | 0 | 46
Participants | 15 | 2 |  | 14

18. Secondary Outcome: Number of Participants With Categorical Change From Baseline to Last Post-Baseline in Sitting Systolic and Diastolic Blood Pressure During Treatment Period
Description: Change categories for sitting systolic blood pressure measured in millimeter of mercury (mm Hg) were as follows: change <=-40, change >-40 to -30, change >-30 to -20, change >-20 to -10, change >-10 to 0, change >0 to <10, change >=10 to <20, change >=20 to <30, change >=30 to <40 and change >=40. Change categories for sitting diastolic blood pressure measured in mm Hg were as follow: change <=-30, change >-30 to -20, change >-20 to -10, change >-10 to 0, change >0 to <10, change >=10 to <20, change >=20 to <30 and change >=30. Rows with only non-zero data/values, for at least 1 reporting arm, are reported below.
Time Frame: Baseline (Day 1, before dosing) up to Week 24
Population: The safety analysis set was defined as all participants treated with tanezumab or placebo SC, including participants who received tanezumab 10 mg prior to protocol amendment 3. Here, "Overall Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 10 mg | Tanezumab 10/20 mg | Tanezumab 20 mg
Number analyzed (Participants) | 67 | 9 | 1 | 68
Participants
  Sitting Systolic Blood Pressure (mmHg) Change <=-40 | 1 | 0 | 0 | 1
  Sitting Systolic Blood Pressure (mmHg) Change >-40 to -30 | 1 | 0 | 0 | 2
  Sitting Systolic Blood Pressure (mmHg) Change >-30 to -20 | 6 | 0 | 1 | 3
  Sitting Systolic Blood Pressure (mmHg) Change >-20 to -10 | 10 | 3 | 0 | 14
  Sitting Systolic Blood Pressure (mmHg) Change >-10 to 0 | 26 | 2 | 0 | 25
  Sitting Systolic Blood Pressure (mmHg) Change >0 to <10 | 12 | 1 | 0 | 9
  Sitting Systolic Blood Pressure (mmHg) Change >=10 to <20 | 6 | 3 | 0 | 10
  Sitting Systolic Blood Pressure (mmHg) Change >=20 to <30 | 5 | 0 | 0 | 3
  Sitting Systolic Blood Pressure (mmHg) Change >=30 to <40 | 0 | 0 | 0 | 1
  Sitting Diastolic Blood Pressure (mmHg) Change >-30 to -20 | 0 | 1 | 0 | 1
  Sitting Diastolic Blood Pressure (mmHg) Change >-20 to -10 | 10 | 1 | 1 | 13
  Sitting Diastolic Blood Pressure (mmHg) Change >-10 to 0 | 39 | 4 | 0 | 26
  Sitting Diastolic Blood Pressure (mmHg) Change >0 to <10 | 11 | 0 | 0 | 18
  Sitting Diastolic Blood Pressure (mmHg) Change >=10 to <20 | 5 | 2 | 0 | 9
  Sitting Diastolic Blood Pressure (mmHg) Change >=20 to <30 | 2 | 1 | 0 | 1

19. Secondary Outcome: Number of Participants With Categorical Summary of Electrocardiogram (ECG) (QTC) Data
Description: Electrocardiogram assessment included QT interval corrected using Fridericia's formula (QTcF), QT interval corrected using Bazett's formula (QTcB), both had following categories: 450<=Value<480 millisecond (msec), 480<=Value<500 msec and Value>=500 msec.
Time Frame: Baseline (Day 1, before dosing) up to Week 24
Population: The safety analysis set was analyzed. Here, "Overall Number of Participants Analyzed" signifies number of participants with post-baseline results evaluated against criteria. In reporting arm "Tanezumab10/20 mg", the participant did not have post-baseline results evaluated against ECG (QTC) criteria, hence was not evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 10 mg | Tanezumab 10/20 mg | Tanezumab 20 mg
Number analyzed (Participants) | 40 | 8 | 0 | 44
Participants
  QTCB Interval 450<=Value<480 | 2 | 1 |  | 6
  QTCB Interval 480<=Value<500 | 0 | 0 |  | 1
  QTCF Interval 450<=Value<480 | 1 | 0 |  | 5

20. Secondary Outcome: Number of Participants With Confirmed Orthostatic Hypotension
Description: Orthostatic hypotension was defined as postural change (supine to standing) that met the following criteria: for systolic blood pressure (BP) less than or equal to (<=) 150 millimeter of mercury (mmHg) (mean supine): reduction in systolic BP >=20 mmHg or reduction in diastolic BP >=10 mmHg at the 1 and/or 3 minute standing BP measurements. For systolic BP greater than (>) 150 mmHg (mean supine): reduction in systolic BP >=30 mmHg or reduction in diastolic BP >=15 mmHg at the 1 and/or 3 minute standing BP measurements. If the 1 minute or 3 minute standing BP in a sequence met the orthostatic hypotension criteria, then that sequence was considered positive. If 2 of 2 or 2 of 3 sequences were positive, then orthostatic hypotension was considered confirmed.
Time Frame: Baseline (Day 1, before dosing), Weeks 8, 16, 24 and 48
Population: The safety analysis set included all subjects treated with tanezumab or placebo SC, including subjects who received tanezumab 10 mg prior to protocol amendment 3. Here, "number analyzed" signifies participants evaluable at specific time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 10 mg | Tanezumab 10/20 mg | Tanezumab 20 mg
Number analyzed (Participants) | 73 | 9 | 1 | 72
Participants
  Baseline | 0 | 0 | 0 | 0
  Week 8: number analyzed (Participants) | 44 | 7 | 1 | 52
  Week 8 | 0 | 0 | 0 | 0
  Week 16: number analyzed (Participants) | 34 | 6 | 0 | 43
  Week 16 | 0 | 0 | 0 | 1
  Week 24: number analyzed (Participants) | 33 | 5 | 0 | 37
  Week 24 | 0 | 0 | 0 | 0
  Week 48: number analyzed (Participants) | 28 | 5 | 0 | 26
  Week 48 | 0 | 0 | 0 | 0

21. Secondary Outcome: Number of Participants With Clinically Significant Findings in Weight Measurement, Counted as an AE
Description: The number of participants with clinically significant findings in weight measurement and were counted as an AE in the study were reported in this outcome measure.
Time Frame: Day 1 of dosing up to maximum of Week 48
Population: The safety analysis set included all subjects treated with tanezumab or placebo SC, including subjects who received tanezumab 10 mg prior to protocol amendment 3.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 10 mg | Tanezumab 10/20 mg | Tanezumab 20 mg
Number analyzed (Participants) | 73 | 9 | 1 | 72
Participants | 2 | 0 | 0 | 2

22. Secondary Outcome: Number of Participants With Abnormal Physical Examination at Screening
Description: Physical examination included assessment of general, head, eyes, ears, nose, neck, thyroid, lungs, heart, abdomen, extremities, skin, throat and other. Investigator judged abnormality in physical examinations.
Time Frame: Screening (up to 37 days prior to Day 1)
Population: The safety analysis set included all subjects treated with tanezumab or placebo SC, including subjects who received tanezumab 10 mg prior to protocol amendment 3. Here, "Overall Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure and "number analyzed" signifies participants evaluable at specific time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 10 mg | Tanezumab 10/20 mg | Tanezumab 20 mg
Number analyzed (Participants) | 72 | 9 | 1 | 72
Participants
  General | 3 | 1 | 0 | 6
  Head | 2 | 1 | 0 | 1
  Eyes | 4 | 1 | 0 | 1
  Ears | 1 | 0 | 0 | 1
  Nose | 0 | 0 | 0 | 0
  Neck | 2 | 1 | 0 | 2
  Thyroid: number analyzed (Participants) | 72 | 9 | 1 | 71
  Thyroid | 2 | 0 | 0 | 0
  Lungs | 5 | 1 | 0 | 3
  Heart | 2 | 2 | 0 | 3
  Abdomen: number analyzed (Participants) | 72 | 9 | 1 | 71
  Abdomen | 2 | 1 | 1 | 5
  Extremities: number analyzed (Participants) | 72 | 9 | 1 | 71
  Extremities | 14 | 0 | 0 | 10
  Skin | 15 | 2 | 0 | 10
  Throat | 3 | 1 | 0 | 2
  Other 1: number analyzed (Participants) | 15 | 5 | 0 | 10
  Other 1 | 9 | 3 |  | 6
  Other 2: number analyzed (Participants) | 7 | 4 | 0 | 6
  Other 2 | 1 | 3 |  | 2
  Other 3: number analyzed (Participants) | 6 | 3 | 0 | 4
  Other 3 | 0 | 1 |  | 0

23. Secondary Outcome: Number of Participants With Individual Adjudicated Joint Safety Outcome/Event
Description: Joint-related safety events resulting in total joint replacement and/or discontinuation from the study as well as adverse events were reviewed by the External Adjudication Committee to confirm the potential events as adjudicated join safety event. In this outcome measure, number of participants with any of the joint safety adjudication outcomes of primary osteonecrosis, rapidly progressive osteoarthritis (OA) (type 1 and type 2), subchondral insufficiency fracture (or SPONK), or pathological fracture were reported. Other adjudication outcomes included normal progression of OA and other joint outcome.
Time Frame: During the study, maximum up to Week 48
Population: The safety analysis set was analyzed. Here, "Overall Number of Participants Analyzed" signifies participants who were analyzed by the Adjudication Committee. In reporting arm, "Tanezumab10/20 mg" the participant did not have potential joint related safety event for analysis by Adjudication Committee.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 10 mg | Tanezumab 10/20 mg | Tanezumab 20 mg
Number analyzed (Participants) | 1 | 1 | 0 | 3
Participants
  Rapidly Progressive OA | 0 | 0 |  | 0
  Rapidly Progressive OA type 1 | 0 | 0 |  | 0
  Rapidly Progressive OA type 2 | 0 | 0 |  | 0
  Primary Osteonecrosis | 0 | 0 |  | 0
  Pathological Fracture | 0 | 0 |  | 2
  Subchondral Insufficiency Fracture | 0 | 0 |  | 0
  Normal Progression of OA | 0 | 0 |  | 0
  Other Joint Outcome | 1 | 1 |  | 1

24. Secondary Outcome: Number of Participants With At Least 1 Total Joint Replacements (TJR)
Description: Number of participants with joint replacement surgery were reported.
Time Frame: During the study, maximum up to Week 48
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 10 mg | Tanezumab 10/20 mg | Tanezumab 20 mg
Number analyzed (Participants) | 73 | 9 | 1 | 72
Participants | 0 | 0 | 0 | 1

25. Secondary Outcome: Number of Participants With Anti-Drug Antibodies (ADA) and Neutralizing Anti-Drug Antibodies (NAb)
Description: Human serum ADA samples were analyzed for the presence or absence of anti-tanezumab antibodies by using a semi quantitative enzyme linked immunosorbent assay (ELISA). Number of participants with presence of anti-tanezumab antibodies and neutralizing anti-drug antibodies are reported.
Time Frame: Baseline (Day 1, before dosing) up to Week 48
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 10 mg | Tanezumab 10/20 mg | Tanezumab 20 mg
Number analyzed (Participants) | 73 | 9 | 1 | 72
Participants
  ADA | 0 | 0 | 0 | 1
  NAb | 0 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: Day 1 of dosing up to 24 weeks post last dose (maximum up to Week 48)
Description: Same event may appear as AE and SAE, what is presented are distinct events. Event may be categorized as serious in 1 participant and as non-serious in another participant or 1 participant may have experienced both serious and non-serious event during study. Safety analysis set was evaluated.
Arm/Group | Placebo | Tanezumab 10 mg | Tanezumab 10/20 mg | Tanezumab 20 mg
All-Cause Mortality (participants affected / at risk) | 23/73 | 1/9 | 1/1 | 21/72
Serious Adverse Events (participants affected / at risk) | 52/73 | 9/9 | 1/1 | 62/72
Other Adverse Events (participants affected / at risk) | 43/73 | 8/9 | 1/1 | 49/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=73) | Tanezumab 10 mg (N=9) | Tanezumab 10/20 mg (N=1) | Tanezumab 20 mg (N=72)
Anaemia (Blood and lymphatic system disorders) | 12 | 1 | 1 | 10
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 3 | 0 | 0 | 2
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 1
Keratitis (Eye disorders) | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 0 | 1
Visual acuity reduced (Eye disorders) | 0 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 3 | 2 | 1 | 6
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 6
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Gingival bleeding (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gingival swelling (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Loose tooth (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 6 | 0 | 0 | 4
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 4 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 6 | 1 | 1 | 4
Application site reaction (General disorders) | 1 | 0 | 0 | 0
Asthenia (General disorders) | 4 | 0 | 1 | 7
Chest pain (General disorders) | 1 | 0 | 0 | 0
Cyst (General disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 5 | 1 | 1 | 6
Feeling cold (General disorders) | 1 | 0 | 0 | 0
Gait disturbance (General disorders) | 1 | 0 | 0 | 0
Inflammation (General disorders) | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 1 | 1 | 0 | 4
Oedema peripheral (General disorders) | 2 | 0 | 0 | 9
Pain (General disorders) | 3 | 0 | 0 | 6
Peripheral swelling (General disorders) | 1 | 0 | 0 | 2
Pyrexia (General disorders) | 2 | 1 | 0 | 2
Swelling (General disorders) | 1 | 0 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Liver injury (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Ocular icterus (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Allergy to plants (Immune system disorders) | 0 | 0 | 0 | 1
Contrast media allergy (Immune system disorders) | 0 | 1 | 0 | 0
Bacterial infection (Infections and infestations) | 0 | 0 | 0 | 2
Body tinea (Infections and infestations) | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 2
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 1
Cystitis (Infections and infestations) | 2 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0
Gingivitis (Infections and infestations) | 1 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 4
Onychomycosis (Infections and infestations) | 0 | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 1 | 0 | 1
Oral fungal infection (Infections and infestations) | 0 | 0 | 0 | 1
Periodontitis (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 3 | 0 | 0 | 4
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0 | 0
Tinea versicolour (Infections and infestations) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 1
Viral infection (Infections and infestations) | 1 | 0 | 0 | 1
Avulsion fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 3 | 0 | 0 | 5
Foot fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Nerve injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 2 | 0 | 0 | 0
Blood creatine phosphokinase decreased (Investigations) | 1 | 0 | 0 | 0
Blood creatinine decreased (Investigations) | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1
Body temperature increased (Investigations) | 1 | 0 | 0 | 1
Carbohydrate antigen 15-3 increased (Investigations) | 1 | 0 | 0 | 0
Carcinoembryonic antigen increased (Investigations) | 1 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0 | 0
Haematology test abnormal (Investigations) | 0 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 1 | 0 | 0 | 0
Neutrophil count increased (Investigations) | 1 | 0 | 0 | 0
Occult blood positive (Investigations) | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0 | 1
Squamous cell carcinoma antigen (Investigations) | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 3 | 0 | 0 | 3
Weight increased (Investigations) | 0 | 1 | 0 | 0
White blood cell count decreased (Investigations) | 2 | 0 | 0 | 0
Acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 4 | 1 | 1 | 10
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 0 | 0 | 0
Hypocholesterolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypophagia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Mineral deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 2 | 0 | 11
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 1 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 0 | 0 | 3
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 3
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Thoracic spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Vertebral osteophyte (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 1 | 0 | 7
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 0 | 2
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 0 | 4
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 3
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Metastases to ovary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 1 | 1 | 9
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Burning sensation (Nervous system disorders) | 0 | 0 | 0 | 1
Cerebrovascular insufficiency (Nervous system disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 3 | 0 | 0 | 3
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 2 | 1 | 0 | 5
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 0 | 0 | 1
Neuralgia (Nervous system disorders) | 2 | 0 | 0 | 2
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 2
Paraparesis (Nervous system disorders) | 1 | 0 | 0 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0
Polyneuropathy (Nervous system disorders) | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1
Radiculopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Sacral radiculopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0 | 0
Sensory disturbance (Nervous system disorders) | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 2 | 1 | 0 | 2
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 0 | 1
Trigeminal neuralgia (Nervous system disorders) | 1 | 0 | 0 | 0
Adjustment disorder with depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 3 | 0 | 0 | 0
Depressed mood (Psychiatric disorders) | 3 | 0 | 1 | 2
Depression (Psychiatric disorders) | 2 | 0 | 0 | 2
Hyposomnia (Psychiatric disorders) | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 1 | 0 | 5
Nervousness (Psychiatric disorders) | 0 | 0 | 0 | 1
Sleep disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 2 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 2
Hypertonic bladder (Renal and urinary disorders) | 0 | 0 | 0 | 1
Micturition disorder (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal cyst (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 2 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 2
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 1
Breast disorder (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Oedema genital (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Sputum retention (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 2
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Onycholysis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 2 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 4 | 0 | 0 | 1
Scab (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin oedema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 2
Hot flush (Vascular disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 0 | 2
Lymphoedema (Vascular disorders) | 2 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 1 | 0 | 1
Pallor (Vascular disorders) | 0 | 0 | 0 | 2
Pelvic venous thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0 | 0 | 0
Peripheral artery aneurysm (Vascular disorders) | 1 | 0 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 0 | 1
Post thrombotic syndrome (Vascular disorders) | 0 | 0 | 0 | 1
Thrombophlebitis (Vascular disorders) | 1 | 0 | 0 | 0
Vascular fragility (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=73) | Tanezumab 10 mg (N=9) | Tanezumab 10/20 mg (N=1) | Tanezumab 20 mg (N=72)
Anaemia (Blood and lymphatic system disorders) | 9 | 1 | 1 | 9
Leukopenia (Blood and lymphatic system disorders) | 3 | 0 | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0
Visual acuity reduced (Eye disorders) | 0 | 1 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 3 | 2 | 1 | 6
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 6
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 6 | 0 | 0 | 4
Toothache (Gastrointestinal disorders) | 4 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 6 | 0 | 1 | 4
Asthenia (General disorders) | 4 | 0 | 1 | 6
Fatigue (General disorders) | 5 | 1 | 1 | 6
Influenza like illness (General disorders) | 1 | 1 | 0 | 4
Oedema peripheral (General disorders) | 2 | 0 | 0 | 9
Pain (General disorders) | 3 | 0 | 0 | 6
Peripheral swelling (General disorders) | 1 | 0 | 0 | 2
Pyrexia (General disorders) | 2 | 0 | 0 | 2
Contrast media allergy (Immune system disorders) | 0 | 1 | 0 | 0
Bacterial infection (Infections and infestations) | 0 | 0 | 0 | 2
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 2
Cystitis (Infections and infestations) | 2 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 4
Oral candidiasis (Infections and infestations) | 0 | 1 | 0 | 11
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 3
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 3 | 0 | 0 | 5
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 2 | 0 | 0 | 0
Weight decreased (Investigations) | 3 | 0 | 0 | 3
Weight increased (Investigations) | 0 | 1 | 0 | 0
White blood cell count decreased (Investigations) | 2 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 4 | 1 | 1 | 10
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 2 | 0 | 11
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 0 | 0 | 3
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0 | 4
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 2
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 3
Dizziness (Nervous system disorders) | 3 | 0 | 0 | 3
Headache (Nervous system disorders) | 2 | 1 | 0 | 5
Neuralgia (Nervous system disorders) | 2 | 0 | 0 | 2
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 2
Somnolence (Nervous system disorders) | 2 | 1 | 0 | 2
Anxiety (Psychiatric disorders) | 3 | 0 | 0 | 0
Depressed mood (Psychiatric disorders) | 3 | 0 | 1 | 2
Depression (Psychiatric disorders) | 2 | 0 | 0 | 2
Insomnia (Psychiatric disorders) | 1 | 1 | 0 | 5
Dysuria (Renal and urinary disorders) | 2 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 2 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 2 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 4 | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 0 | 2
Lymphoedema (Vascular disorders) | 2 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 1 | 0 | 1
Pallor (Vascular disorders) | 0 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2018-06-14): https://cdn.clinicaltrials.gov/large-docs/28/NCT02609828/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-08): https://cdn.clinicaltrials.gov/large-docs/28/NCT02609828/SAP_001.pdf